Effects of teriparatide and risedronate on new fractures in post-menopausal women with severe osteoporosis (VERO): a multicentre, double-blind, double-dummy, randomised controlled trial (VERtebral fracture treatment comparisons in Osteoporotic women, VERO trial)

**DUPLICATE VERO** 

April 30, 2021

NCT01709110

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Effects of teriparatide and risedronate on new fractures in post-menopausal women with severe osteoporosis (VERO): a multicentre, double-blind, double-dummy, randomised controlled trial (<u>VERtebral fracture treatment comparisons in Osteoporotic women, VERO trial - NCT01709110</u>)

#### 1.2 Intended aim(s)

To assess the effects of 24 months of treatment with teriparatide compared with risedronate on the incidence of new fractures in post-menopausal women with preexisting vertebral fractures, regardless of previous osteoporosis treatment.

### 1.3 Primary endpoint for replication

New vertebral fracture.

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming a 24-month new vertebral fracture incidence of 4.5% in the teriparatide group and 10% in the risedronate group, 466 patients per group would provide 90% power to detect a difference between groups in the incidence of new vertebral fractures using a Pearson  $\chi^2$  test (two-sided  $\alpha$  of 0.05).

### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Non-vertebral fracture.

#### 1.6 <u>Trial estimate</u>

Hazard Ratio, HR = 0.44 (95% CI, 0.29 to 0.68) comparing teriparatide vs. risedronate group during a 24-month period (Kendler et al., 2007).

## 2. Person responsible for implementation of replication in Aetion

Elvira D'Andrea, MD, MPH, implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum CDM, IBM® MarketScan®

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1. Design Diagram – VERO TRIAL REPLICATION



#### 5. Cohort Identification

### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing injectable subcutaneous teriparatide (20 µg daily) to oral risedronate (35 mg weekly). The patients will be required to have continuous enrollment during a baseline period of 365 days before initiation of teriparatide or oral risedronate. We will restrict the analyses to women older than 45 with osteoporosis and history of vertebral fractures.

### 5.2 Important steps for cohort formation

New use of teriparatide (exposure) is defined as no use of the exposure drug within the 730 days (2 years) prior to index date. This will emulate the trial requirement for which treatment with teriparatide was not allowed any time before randomization. New use of risedronate (comparator) is defined as no use of the comparator drug within the 180 days prior to index date. The shorter washout period for risedronate users, compared to teriparatide users, will emulate the trial requirement of discontinuation of risedronate at the beginning of the screening period. Differently from teriparatide, history of risedronate use was allowed in the trial. New users of teriparatide are not allowed to receive risedronate within the 180 days prior to index date, and new users of risedronate are not allowed to receive teriparatide within the 730 days (2 years) prior to index date.

#### 5.2.1 Eligible cohort entry dates

Teriparatide indication for treatment of osteoporosis in postmenopausal women was approved by FDA on Nov 26, 2002 (the approval of risedronate for the same indication was antecedent to 2002). The initial eligible cohort entry date was the first date after Nov 26, 2002 commonly available in both the databases investigated (IBM® MarketScan®, Optum CDM). The last date eligible as cohort entry date was the end of available data for IBM® MarketScan®. For Optum CDM, we excluded the data cut that overlaps with the COVID-19 pandemic (range: April 1st - Jun 30th, 2020), since we assumed a higher proportion of drug discontinuation in that time period. The following eligible cohort entry dates were included:

- IBM® MarketScan®: Jan 1, 2004 (start of available data) December 31, 2018 (end of available data)
- Optum CDM: Jan 1, 2004 (start of available data) Mar 31, 2020
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.
- 5.3 Flowchart of the study cohort assembly

For teriparatide vs. risedronate

| | Optum CDM | | IBM® Mai | ·ketScan® |
|---|---|---|---|---|
| | Excluded Patients | Remaining<br>Patients | Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78202636 | | 200203908 |
| Did not meet cohort entry criteria | -77830806 | 371830 | -199450502 | 753406 |
| Excluded due to insufficient enrollment | -90897 | 280933 | -176733 | 576673 |
| Excluded due to prior use of referent | -199055 | 81878 | -403827 | 172846 |
| Excluded due to prior use of exposure | -19897 | 61981 | -44254 | 128592 |
| Excluded because patient qualified in >1 exposure category | 0 | 61981 | 0 | 128592 |
| Excluded based on Inclusion criteria #1 - Age >= 45 | -1814 | 60167 | -3865 | 124727 |
| Excluded based on Inclusion criteria #2 - Female | -4439 | 55728 | -9140 | 115587 |
| Excluded based on Inclusion criteria #3.1 - History of vertebral fracture (including from inception to 90 days) | -48548 | 7180 | -103348 | 12239 |
| Excluded based on Inclusion criteria #3.2 - Vertebral fracture diagnosis excluded in the 90 days before cohort entry | -740 | 6440 | -969 | 11270 |
| Excluded based on Inclusion criteria #4 - Osteoporosis | -3 | 6437 | -18 | 11252 |
| Excluded based on Exclusion criteria #1 - Pregnancy | -1 | 6436 | -1 | 11251 |
| Excluded based on Exclusion criteria #2 - Paget's Disease | -5 | 6431 | -9 | 11242 |
| Excluded based on Exclusion criteria #3.1 - Renal Osteodystrophy | -2 | 6429 | -1 | 11241 |
| Excluded based on Exclusion criteria #3.2 - Osteomalacia | -11 | 6418 | -12 | 11229 |
| Excluded based on Exclusion criteria #3.3 - Cushing syndrome and other disorders of adrenal glands | -35 | 6383 | -62 | 11167 |
| Excluded based on Exclusion criteria #3.4 - Hyperparathyroidism and hypoparathyroidism | -60 | 6323 | -86 | 11081 |
| Excluded based on Exclusion criteria #3.5 - Intestinal malabsorption | -27 | 6296 | -41 | 11040 |
| Excluded based on Exclusion criteria #4 - Hypercalcemia and Hypocalcemia | -14 | 6282 | -23 | 11017 |
| Excluded based on Exclusion criteria #5 - Malignant neoplasm, excluding non-melanoma skin cancer | -500 | 5782 | -936 | 10081 |
| Excluded based on Exclusion criteria #6 - End-stage liver disease (ESLD) | -31 | 5751 | -51 | 10030 |
| Excluded based on Exclusion criteria #7 – End-stage renal disease (ESRD) | -6 | 5745 | -14 | 10016 |
| Excluded based on Exclusion criteria #8 - Nephrolithiasis or urolithiasis | -52 | 5693 | -109 | 9907 |
| Excluded based on Exclusion criteria #9 - Kyphoplasty or vertebroplasty | -17 | 5676 | -47 | 9860 |

| Excluded based on Exclusion criteria #10 - Osteonecrosis of the jaw | 0 | 5676 | -2 | 9858 |
|---|---|---|---|---|
| Excluded based on Exclusion criteria #11 - Atypical subtrochanteric or diaphyseal femoral fractures | -28 | 5648 | -55 | 9803 |
| Excluded based on Exclusion criteria #12 - Upper gastrointestinal disorders | -170 | 5478 | -221 | 9582 |
| Excluded based on Exclusion criteria #13 - CCI (180 days) | -2 | 5476 | -1 | 9581 |
| Excluded based on Exclusion criteria #14 - Drug addiction or alcohol abuse or not compliant | -91 | 5385 | -58 | 9523 |
| Excluded based on Exclusion criteria #15 - Oral bisphosphonate use | -499 | 4886 | -1024 | 8499 |
| Excluded based on Exclusion criteria #16 - SERMs, Calcitonin, HRT | -101 | 4785 | -321 | 8178 |
| Excluded based on Exclusion criteria #17 - Zoledronic acid use | -2 | 4783 | -7 | 8171 |
| Excluded based on Exclusion criteria #18 - Intravenous ibandronate or pamidronate | -1 | 4782 | -1 | 8170 |
| Excluded based on Exclusion criteria #19 - Denosumab use | -10 | 4772 | -4 | 8166 |
| Excluded based on Exclusion criteria #20 - PTH or PTH analogue use | -44 | 4728 | -137 | 8029 |
| Excluded based on Exclusion criteria #21 - Romosozumab | 0 | 4728 | 0 | 8029 |
| Final cohort | | 4728 | | 8029 |

#### 6. Variables

# 6.1 Exposure-related variables:

#### Study drug:

New initiation of injectable subcutaneous teriparatide (20 µg daily). New initiation is defined as no use of teriparatide in the prior 730 days before treatment initiation (washout period). New users of teriparatide are not allowed to receive risedronate within the 180 days prior to treatment initiation.

### Comparator agent:

New initiation of oral risedronate (35 mg weekly). New initiation is defined as no use of risedronate in the prior 180 days before treatment initiation (washout period). New users of risedronate are not allowed to receive teriparatide within the 730 days prior to treatment initiation.

## 6.2 <u>Preliminary Covariates:</u>

- Age
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and

including index date.

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**). Gender is not included since the study is already restricted to female subjects.

## 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- **Primary outcome:** Vertebral fracture (algorithm adapted from Wright et al. 2019)
- Secondary outcome: Non-vertebral fracture

### 6.3.2 Study follow-up

As-treat (AT) analysis will be conducted with treatment defined as the index drug on the day of cohort entry. Similar to the trial, the patients will be followed for 24 months. A grace period and a risk exposure window of 60 days will be considered in the primary analysis.

The follow-up will start the day after drug initiation (i.e., cohort entry date), as described in the VERO trial, and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continuous registration in the database,
- Discontinuation of the index drugs,
- Addition of the index drug from the other group or crossover,
- End of the study period,
- Measured death event occurs,
- Nursing home admission

 Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.

A subgroup analysis will be performed by age categorized by tertiles () emulating one of the prespecified subgroup analyses of the VERO trial (Geusens P et al. 2018).

### 7. Initial Feasibility Analysis

# Action report name:

For teriparatide vs. risedronate

Optum CDM - https://bwh-dope.aetion.com/projects/details/1640/results/66361/result/0

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1641/results/66364/result/0

Date conducted: 02/25/2021

Complete Aetion feasibility analysis using age and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population FEASIBILITY- FOR STUDY OUTCOME
- Report reasons for censoring in the overall study population
- Report overall risk of the primary outcome.

#### 8. Initial Power Assessment

#### Aetion report name:

For teriparatide vs. risedronate

Optum CDM - https://bwh-dope.aetion.com/projects/details/1640/results/66362/result/0

IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1641/results/66363/result/0

Date conducted: 02/25/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 2 covariates: age and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 03/17/2021 |
|-------------------------|------------------|----------------|------------|
| | Jessica Franklin | | |
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 03/16/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

For teriparatide vs. risedronate

Optum CDM: https://bwh-dope.aetion.com/projects/details/1640/rwrs/67726

IBM® MarketScan®: https://bwh-dope.aetion.com/projects/details/1641/rwrs/67727

Date conducted: 03/29/21

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0%) | 0 (0%) | 0 (0%) |
| Death | 28 (0.65%) | 9 (0.21%) | 19 (0.44%) |
| End of patient enrollment | 715 (16.5%) | 300 (6.92%) | 415 (9.58%) |
| End of index exposure | 157 (3.62%) | 70 (1.62%) | 87 (2.01%) |
| Maximum follow-up time | 442 (10.20%) | 185 (4.27%) | 257 (5.93%) |
| End of index exposure | 2775 (64.03%) | 1522 (35.12%) | 1253 (28.91%) |
| Start of an additional exposure | 37 (0.85%) | 9 (0.21%) | 28 (0.65%) |
| Nursing Home | 180 (4.15%) | 72 (1.66%) | 108 (2.49%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® | | |
| Overall Patient Population | 163.5 [88 - 415] | 190 [100 - 431.5] |
| Referent - Risedronate | 148 [88 - 371] | 148 [88 - 331] |
| Exposure - Teriparatide | 192 [88 - 446] | 234 [113 - 533] |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | Pooled |
|-------------------------|-----------|------------------|--------|
| Risk per 1,000 patients | 15.9 | 18.9 | 17.8 |

## 10. Final Power Assessment

## Date conducted:

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

### o Pooled

| 0 <u>1 001<b>cu</b></u> | |
|----------------------------|-------------|
| Superiority Analysis | |
| Number of patients matched | 4,334 |
| Reference | 2,167 |
| Exposed | 2,167 |
| Risk per 1,000 patients | 17.80 |
| Desired HR from RCT | 0.44 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 77.1452 |
| Power | 0.950063363 |

## Optum CDM

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 1,494 |
| Reference | 747 |
| Exposed | 747 |
| Risk per 1,000 patients | 15.90 |
| Desired HR from RCT | 0.44 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 23.7546 |
| Power | 0.516274582 |

# o <u>IBM® MarketScan®</u>

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 2,840 |
| Reference | 1,420 |
| Exposed | 1,420 |
| Risk per 1,000 patients | 18.90 |
| Desired HR from RCT | 0.44 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 53.676 |
| Power | 0.852553869 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 04/16/2021 |
|-------------------------|--------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 04/15/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

# 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns:

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 12. Register study protocol on clinicalTrials.gov

Date conducted: 04/30/2021

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Action report name:

Date conducted:

### 13.1 <u>For primary analysis</u>:

# 13.2 For sensitivity analyses:

# 14. Requested Results

# 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | le Before adjustment | | After adjust | ment | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |
| ••• | | | | | | |

# 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| Overall | Referent | Exposure |
|---------|----------|----------|
|---------|----------|----------|

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Outcome |
|---------------------------------|
| Death |
| Start of an additional exposure |
| End of index exposure |
| Specified date reached |
| End of patient data |
| End of patient enrollment |

# 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |
| ••• | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

# 14.5 <u>Table 5: Results from secondary analyses.</u>

#### 15. References

Kendler DL, Marin F, Zerbini CAF, Russo LA, Greenspan SL, Zikan V, Bagur A, Malouf-Sierra J, Lakatos P, Fahrleitner-Pammer A, Lespessailles E, Minisola S, Body JJ, Geusens P, Möricke R, López-Romero P. Effects of teriparatide and risedronate on new fractures in post-menopausal women with severe osteoporosis (VERO): a multicentre, double-blind, double-dummy, randomised controlled trial. *Lancet*. 2018 Jan 20;391(10117):230-240. doi: 10.1016/S0140-6736(17)32137-2.

Wright NC, Daigle SG, Melton ME, Delzell ES, Balasubramanian A, Curtis JR. The Design and Validation of a New Algorithm to Identify Incident Fractures in Administrative Claims Data. *J Bone Miner Res.* 2019 Oct;34(10):1798-1807. doi: 10.1002/jbmr.3807.

Geusens P, Marin F, Kendler DL, Russo LA, Zerbini CA, Minisola S, Body JJ, Lespessailles E, Greenspan SL, Bagur A, Stepan JJ, Lakatos P, Casado E, Moericke R, López-Romero P, Fahrleitner-Pammer A. Effects of Teriparatide Compared with Risedronate on the Risk of Fractures in Subgroups of Postmenopausal Women with Severe Osteoporosis: The VERO Trial. *J Bone Miner Res.* 2018 May;33(5):783-794. doi: 10.1002/jbmr.3384.

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177.

| # | VERO trial definitions | Implementation in routine care | | gle Drive for further details or any missing information: ilders/IWD618wnywYiEaXzfl.TcuK-VCcnb6b-gV?usp=sharing |
|---|---|---|---|---|
| | Trial details - clinicaltr | ial.gov NCT01709110 | lists will be available in the above Google Drive Fold<br>macro that implements forward/ba | excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code<br>or [link above]. ICD-9 to ICD-10 code conversions were completed using a SAS<br>sckward mapping based on the CMS ICD-9 to ICD-10 mapping:<br>1-10-cm-and-pc-sc-rosswalk-general-equivalence-mapping.html |
| | EXPOSURE vs. | COMPARISON | References/Rationale | Color coding |
| | | Exposure: new use of Teriparatide (washout 730 days) | | |
| | | NDC Generic Name: TERIPARATIDE | | |
| E | Exposure: 20 µg ofteriparatide once daily | NDC codes: 00002897101, 54868540600, 00002840001, 47781065289 | Washout period - Criteria 20.1, 20.7 | Criteria |
| | | Brand names: FORTEO | | |
| | | CPT/HCPCS Procedure Code: J3110 | | |
| | | Comparator: new-use of Risedronate (washout 180 days) | | |
| | | NDC Generic Name: RISEDRONATE SODIUM, RISEDRONATE SODIUM/CALCIUM CARBONATE | | |
| c | Reference: 35 mg of oral risedronate once weekly Aim: To compare the anti-fracture efficacy of teriparatide with risedronate in patients with severe osteoporosis | NDC codes: 00093309819, 00093309829, 00093309844, 00093309956, 00093310056, 00093550919, 00093550944, 00093777113, 00093777119, 00093777119, 00149047201, 01149047201, 01149047201, 00149047201, 00149047201, 00149047201, 00149047501, 00149047701, 00149047801, 0014904 | | Adequate mapping in claims |
| | | Brand names: ACTONEL, ATELVIA | | |
| | PRIMARY | DUTCOME Measured 1 day after drug initiation: | | Intermediate mapping in claims |
| | New radiographic vertebral fractures during a 24-month study period. [Lateral spine radiographs were repeated at 12 and 24 months or early termination for new vertebral fractures. Additional unscheduled radiographs were done at any interim visit to detect new clinical vertebral fractures if the patient reported back pain clinically suggestive of a vertebral fracture.] | Vertebral Fractures: Algorithm include the following case-qualifying (CQ): CQ = 1 Inpatient claim with primary diagnosis code (ICD9 dx: 805.x, 806.x, 733.13 (ICD10 dx: 512.0xxx,512.0xx85-512.6xxx, 512.6xx8, 512.522.0xx8, 522.0xx8 (excluding "traumatic" and "burst" fractures which are high-energy fractures), M48.50XA, M80.08XA (excluding "stress" and "fatigue" fractures which are fractures caused by abnormal stress on normal bones) OR CQ = 2 Non-inpatient claim with any diagnosis code [ICD9 dx: 805.x, 806.x, 733.13; ICD10 dx: 512.0xxA, 512.0xx8, 51 | Wright NC, Daigle SG, Melton ME, Delzell ES, Balasubramanian A, Curtis JR. The Design and Validation of a New Algorithm to Identify Incident Fractures in Administrative Claims Data. J Bone Miner Res. 2019 Cct;34(10):1798-1807. doi:10.1002/jbmr.3807. Epub 2019 Aug 5. PMID: 31170317. | Poor mapping or cannot be measured in claims |
| | INCLUSION | CRITERIA | | Can't be measured in claims but not important for the analysis |
| 1 | Postmenopausal women ≥ 45 years of age at the time of entry into the trial, whose last menstrual period occurred at least 2 years prior to entry into the trial, and are sufficiently mobile to complete study visits. | Female, ≥ 45 years of age at the time of drug initiation | | |
| 2 | Women < 55 years of age in whom a bilateral oophorectomy cannot clearly be documented must have their postmenopausal status confirmed by a serum FSH level > 40 IU/L and serum estradiol level < 20 pg/mL or < 73 pmol/L. | Measured 180 days prior to and including day of drug initiation in inpatient or outpatient care setting (any diagnosis position): | | |
| 1 | | Excluded if patients had pregnancy codes Pregnancy (see "Pregnancy codes") | | |

| ı | | <u> </u> | |
|---|---|---|---|
| 2 | Aminimum of 2 moderate (SQ2) or 1 severe (SQ3) vertebral fragility fractures [radiographic evidence of at least two moderate (ie, a reduction in vertebral body height of 26–40%) or one severe (more than 40% reduction) prevalent vertebral fragility fracture) | Measured from enoriment to 90 days prior to the day of drug initiation in inpatient or outpatient care setting (any position): Vertebral Fractures diagnosis: ICDS diagnosis codes: M84.4, M84.5, M80.x, S12.x, S22.x, S32.x Vertebral fracture procedures: HCPCS codes: 22305, 22310, 22315, 22318, 22319, 22325-22328, 22510-22515, 22520-22525, 27200, 27202, 72291, 72292, 76012, 76013, 77082, 77085, 73260-52363 ICD10 px: D073xx, D074xx, OPR3xx, OPR4xx, OPS3xx, OPS4xx ICD-9 px: 03.53 | NB. We excluded patients with diagnosis of vertebral fractures from 89 days prior to and including the day of drug initiation to increase the probability of measuring incident vertebral fractures and not prevalent vertebral fractures. The 90-day gap is described in: Wright NC, Daigle SG, Melton ME, Delzell ES, Balssubramanian A, Curtis JR. The Design and Validation of a New Algorithm to Identify Incident Fractures in Administrative Claims Data. J Bone Miner Res. 2019 Oct;34(10):1798-1807. doi: 10.1002/jbmr.3807. |
| 3 | AP lumbar spine or total hip or femoral neck BMD ≥ 1.5 SD below the average BMD for young healthy, non-Hispanic, Caucasian women (T-score ≤ −1.5 SD). | Measured start of all available data and including day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Osteoprosis diagnosis (ICD-9 diagnosis: 733.00, 733.01, 733.02, 733.03, 733.09, 733.13 (ICD-9 diagnosis: M81.0, M81.6, M81.8, M80.88*, M80.00*, M80.01*, M80.02*, M80.03*, M80.04*, M80.05*, M80.06*, M80.07*, M80.08* OR Osteoprosis treatments: Alendronate, Ibandronate, Risedronate, Etidronate, Tiludronate, Denosumab, Calcitonin, Romosozumab, Raloxifene, ZA, Pamidronate (reported as osteoprosis drug in the VERO trial) | |
| 4 | Without language barrier, cooperative, able to come to the clinic for all follow-up visits; has given informed consent before entering the study and after being informed of the medications and procedures to be used in this study. | N/A | |
| 5 | In the opinion of the investigator, is willing to be trained and to use the pen injector daily, is able to satisfactorily use a pen-type injection delivery system, or is willing to receive daily subcutaneous injections from a caregiver who has been trained to use the pen injector. | N/A | |
| | EXCLUSION | NCRITERIA | |
| 1.1 | increased baseline risk of osteosarcoma. This includes patients with Paget's disease of the bone []. As elevation of serum alkaline phosphatase activity may indicate the presence of Paget's disease, an unexplained elevation of this enzyme activity will also be exclusionary. | Measured 365 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): ICD-9 diagnosis: 731.0 Osteitis deformans without mention of bone tumor (Paget's Disease) ICD-10 diagnosis: M88.xxx Osteitis deformans [Paget's disease of bone] + Tiludronate (exclusion criteria 21.1) | |
| 1.2 | [] previous primary skeletal malignancy, or skeletal exposure to therapeutic irradiation. | Captured in criteria 13 | |
| 2 | History of unresolved skeletal diseases that affect bone metabolism, other than osteoporosis, including renal osteodystrophy, osteomalacia, hyperparathyroidism (uncorrected), hypoparathyroidism, and intestinal malabsorption. | Measured 365 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Renal osteodystrophy ICD-9 diagnosis: 588.0 ICD-10 diagnosis: NS5.0 Osteomalacia ICD-9 diagnosis: NS5.0 Osteomalacia ICD-9 diagnosis: NS3.x Cushing syndrome and disorders of adrenal glands: ICD-9 diagnosis: 255.xx ICD-10 diagnosis: E24.x Hyperacrathyroidism and hypoparathyroidism: ICD-9 diagnosis: 252.x, S88.81 ICD-10 diagnosis: 252.x, S88.81 ICD-10 diagnosis: PS5.xx ICD-9 diagnosis: PS5.xx ICD-9 diagnosis: S79.xx ICD-9 diagnosis: C21.x S88.81 Intestinal Malabsorption: Cellac disease, Tropical sprue, Pancreatic steatorrhea, Non-cellac gluten sensitivity, Malabsorption due to intolerance elsewhere classified. Whitoles disease. Other intestinal malabsorption: ICD-9 diagnosis: S79.xx, 040.2 ICD-10 diagnosis: K90.xx | |
| 3 | Abnormally elevated values of serum albumin-corrected calcium levels at baseline, defined as $\geq 10.6$ mg/dL (or $\geq 2.65$ mmol/L). In cases with borderline non-eligible values ( $\geq 10.6$ and $\leq 10.7$ mg/dL), a re-test would be allowed during the screening period. | Measured 30 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Hypercalcemia and Hypocalcemia. ICD-9 diagnosis: 275.41, 275.42 ICD-10 diagnosis: E83.51, E83.52 | |
| 4 | Abnormally low values of serum albumin-corrected calcium levels at baseline, defined as < 8.0 mg/dL (or < 2.0 mmol/L).<br>In cases with borderline non-eligible values (> 7.8 to < 8.0 mg/dL), a retest would be allowed during the screening<br>period to allow normalization with vitamin D and calcium supplements before the randomization visit. | see Criteria 3 | |

# Appendix A

| 5 | Abnormally elevated values of serum intact PTH(1-84) at baseline defined as > 72 pg/mL (or > 7.6 pmol/L). In cases with borderline non-eligible values (> 72 and < 79 pg/mL), a re-test would be allowed during the screening period to allow normalization with vitamin D and calcium supplements before the randomization visit. | see Criteria 2, 3 and 6 |
|---|---|---|
| 6 | Severe vitamin D deficiency at baseline defined as 25-hydroxy-vitamin D levels < 9.2 ng/mL (or < 23 nmol/L). In cases with borderline non-eligible values (> 8.0 and < 9.2 ng/mL), a re-test would be allowed during the screening period to allow normalization with vitamin D supplement before the randomization visit. | N/A |
| 7 | Abnormal thyroid function not corrected by therapy. Patients with subclinical hyperthyroidism or hypothyroidism, defined as abnormally low or high TSH values respectively, with normal fT4 values are eligible to participate in the study. | N/A |
| 8 | History of malignant neoplasms in the 5 years prior to Visit 2, with the exception of superficial basal cell or squamous cell carcinomas of the skin that have been definitively treated. Patients with carcinoma in situ of the uterine cervix treated definitively more than 1 year prior to entry into the study may be randomized. Patients with multiple myeloma or metastases to bone are excluded. | Measured 1825 days (5 years) prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Malignant neoplasm: ICD-9 diagnosis: 140.xx-208.xx (except 173.xx, non-melanoma skin cancer) ICD-10 diagnosis: C00-C43, C45-C97, D45 |
| 9 | Active liver disease or clinical jaundice. Significantly impaired hepatic function, defined as aspartate aminotransferase (AST) > 75 U/L or gamma-glutamyl transpeptidase (GGT) > 300 U/L. | Measured 365 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Cirrhosis: ICD-9 Diagnosis: \$71.2, \$71.5, \$71.6 ICD-10 Diagnosis: \$70.11, K70.2, K70.3x, K70.4x, K74.x Hepatic decompensation: ICD-9 Diagnosis: 456.0, 456.20, 456.1, 456.21, 789.5, 789.59, 572.2, 567.0, 567.2, 567.21, 567.22, 567.29, 567.8, 567.89, 567.9, \$72.4 ICD-10 Diagnosis: R18.x, I85.x, K72.x, K65.x, K66.x, K67 HCC is already excluded with exclusion criteria 13 |
| 10 | Significantly impaired renal function as defined by a calculated endogenous creatinine clearance (CICr) < 30 mL/min using the following Cockcroft-Gault formula for CICr (Cockcroft and Gold 1976) | Measured 365 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Chronic kidnew disease stages IV-V. FSRD 2 codes for occurrence of ESRD/dialysis (either inpatient or outpatient), separated by at least 30 days: ICD-9 Diagnosis: 585.6, V45.1, V56.0, V56.8, S85.5 ICD-9 Procedure: 39.95, 54.98 ICD-10 Diagnosis: 181.5, N18.6, Z49.31, Z49.32, Z99.2 ICD-10 Procedure: 31.95, S4.08 ICD-10 Procedure: 31.95, S4.08 ICD-10 Procedure: 31.95, S4.08 ICD-10 Procedure: 31.95, S4.08 ICD-10 Procedure: 31.95, S4.09.21, S40.002, S41.002, S41 |
| 11 | History of nephrolithiasis or urolithiasis within 1 year prior to Visit 2. | Measured 365 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): ICD-9 Diagnosis: \$92.xx, 274.11 ICD-10 Diagnosis: \$120.xx*\\$23.xx ICD-9 Pix: \$7.0, \$9.95, \$6.0, 98.19, 98.51 ICD-10 Pix: \$7.0, \$9.95, \$6.0, 98.19, 98.51 ICD-10 Pix: OTCB72Z, OTCB8ZZ, OTFB0ZZ, OTFB0ZZ, OTFB4ZZ, OTFB7ZZ, OTFB8ZZ, OTFC0ZZ, OTFC3ZZ, OTFC4ZZ, OTFC7ZZ, OTC8ZZ, OTG97ZZ, OTG98ZZ, OTG7ZZ, OTG8ZZ, OTG7ZZ, OTG8ZZ, OTG7ZZ, OTG8ZZ, OTG7ZZ, OTC8ZZ, OTC7ZZ, OTC8ZZ, OTC7ZZ, OTC8ZZ, OTC7ZZ, OTC8ZZ, OTC8ZZ, OTC7ZZ, OTC8ZZ, OTC8Z |
| 12 | Considered imminent candidates for kyphoplasty or vertebroplasty before Visit 2. | N/A |
| 13 | Patients who have been treated with kyphoplasty or vertebroplasty at 3 or more levels before Visit 2, regardless of the time since the last procedure. | see Criteria 14 |
| 14 | Patients who have been treated with kyphoplasty or vertebroplasty within the last 6 months before Visit 2. | Measured 180 days prior to and including the day of drug initiation in inpatient or outpatient care setting (any diagnosis position): ICD-9 Procedure: Kyphoplasty, 81.66 Vertebroplasty, 81.65 Kyphoplasty, 0813272, OPU3312, OPU3312, OPU3312, OQS0322, OQU0312, OQS1322, OQS13120, OQSS322, OQUS312 Kyphoplasty 0PS3322, OPU3312, OPU3312, OPU4312, OQU0312, OQU0412, OQU1312, OQU1412 CPT: 22514, 22515, 22520, 22521, 22522, 22523, 22524, 22525, O2007, C9718, C9719, S2362, S2363 |

# Appendix A

| | | Measured start of all available data and including day of drug initiation in inpatient or outpatient care setting (any diagnosis | |
|---|---|---|---|
| 15 | Patients with history of osteonecrosis of the jaw or who are, according to the clinical judgment of the investigator, at high risk to develop osteonecrosis of the jaw, including poor oral hygiene, scheduled invasive dental procedures, high doses of bisphosphonates and/or chemotherapy to treat malignancy. | position): History of osteonecrosis of the jaw: ICD-9 diagnosis: 733.45 ICD-10 diagnosis: M87.180 | |
| 16 | Patients with history of atypical subtrochanteric or diaphyseal femoral fractures, according to the diagnostic criteria of the American Society for Bone and Mineral Research Task Force (Shane et al. 2010). | Measured start of all available data and including day of drug initiation in inpatient or outpatient care setting (any diagnosis position): ICD-9 diagnosis: 733.15, 821.0x, 821.1x ICD-10 diagnosis: M84.75, 572.3x | |
| 17 | Active or recent history of significant upper gastrointestinal disorders, such as esophageal disorders which delay esophageal transit or emptying (e.g. stricture or achalasia). | Measured 365 days prior to and including day of drug initiation in inpatient or outpatient care setting (any diagnosis position): ICD-9 diagnosis: \$50.x ICD-10 diagnosis: \$22.x | |
| 18 | Unable to stand or sit in the upright position for at least 30 minutes. | N/A | |
| 19 | Poor medical or psychiatric condition for participating in a clinical study, in the opinion of the investigator. | Measured on the day of drug initiation: CCI >=10 (life expectancy less than the expected duration of the trial) | |
| 20 | History of excessive consumption of alcohol or abuse of drugs in the 1 year prior to Visit 2, in the opinion of the investigator. | Measured 365 days prior to and including day of drug initiation in inpatient or outpatient care setting (any diagnosis position): Alcohol Abuse or Dependence ICD-9 diagnosis: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x (CMS has not released mapping for new ICD10 for this code), V11.3x ICD-10 diagnosis: F10.x, K70.x, G62.1, I42.6, 099.31x OR Prug Abuse or Dependence ICD-9 diagnosis: 292.xx, 304.xx, 305.2x-305.9x, 648.3x ICD-10 diagnosis: F11.x, F12.x, F13.x, F14.x, F15.x, F16.x, F17.2x, F18.x, F19.x, F55.2, G62.0, 099.32x OR Non-compliance: ICD-9 diagnosis: V45.12, V15.81 ICD-10 diagnosis: V45.12, V15.81 ICD-10 diagnosis: V45.12, V15.81 ICD-10 diagnosis: V45.12, V15.81 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagilificin versus other non-gillfozin antidiabetic drugs: population based cohort study." BMJ 2018;360:Xt19 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empaglifiozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empaglifiozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 21.1 | Previous treatment with the following bone active drugs is allowed but treatment must be discontinued at Visit 1 or at the time indicated below: 1. Oral bisphosphonates (including alendronate, risedronate, ibandronate, etidronate). | Measured 180 days prior to and 1 day before the day of drug initiation: <u>Generic names:</u> Alendronate, Ibandronate, Risedronate, Etidronate, Tiludronate | |
| 21.2 | <ol><li>SERMs, calcitonin, estrogen (oral, transdermal, or injectable), progestin, estrogen analog, estrogen agonist, estrogen<br/>antagonist or tibolone, androgens, strontium ranelate, or active vitamin D3 analogues.</li></ol> | Measured 30 days prior to and 1 day before the day of drug initiation: Generic names: SERMS: OSPEMIFENE, RALOXIFENE HCL, ESTROGENS, CONJUGATED/BAZEDOXIFENE ACETATE Calcitonin HRT: estrogens, progestins, androgens | Strontium not approved in USA for treatment of osteoporosis. Vitamin D3 analogues over the counter |
| 21.3 | Intravenous zoledronate, if the last dose was administered at least 12 months before Visit 1. | Measured 365 days prior to and 1 day before the day of drug initiation: Seneric name: Zoledronic Acid Soledronic A | |
| 21.4 | Intravenous ibandronate or pamidronate, if the last dose was administered at least 3 months before Visit 1. | Measured 90 days prior to and 1 day before the day of drug initiation: <u>Generic name</u> ; Ibandronate or pamidronate <u>CPT codes</u> ; C9229, J1740, C9411, J2430 | |
| 21.5 | Subcutaneous denosumab, if the last dose was administered at least 6 months before Visit 1. | Measured 180 days prior to and 1 day before the day of drug initiation: <u>Generic name</u> , Denosumab | |
| 21.6 | Fluoride unless given at therapeutic doses (> 20 mg/day) for more than 3 months in the 2 years prior to Visit 1, or for more than a total of 2 years, or at any dosages within the 6 months prior to Visit 2 (previous or current use of fluoridated water or topical dental fluoride treatment is permitted). | N/A | Sodium Fluoride is not used to treat the osteoporosiss since 2001/2002 when a RCT and sub meta-analysis showed an increased of risk of fractures in the exp arm |
| 21.7 | Prior treatment with PTH, teriparatide, or other PTH analogs; or prior participation in any other clinical trial studying PTH, teriparatide, or other PTH analogs. | Measured 730 days (2 years) prior to and 1 day before the day of drug initiation: Generic names: parathyroid hormone, teriparatide, abaloparatide | |
| 22 | Known hypersensitivity to teriparatide or risedronate, or to any diluents or excipients of teriparatide or risedronate 35 mg/week oral tablet. | N/A | |

# Appendix A

| 23 | Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. | |
|---|---|---|
| | Site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted. | N/A |
| 25 | Lilly employees or employees of third-party organizations (TPOs) involved in study who require exclusion of their employees. | N/A |
| 26 | Romosozumab | Measured 180 days prior to and 1 day before the day of drug initiation: Generic name: Romosozumab Generic name: |

## Pregnancy Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION 72.4 FORCEPS ROTATION OF FETAL HEAD 72.5 BREECH EXTRACTION 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD 72.52 OTHER PARTIAL BREECH EXTRACTION

72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD

72.54 OTHER TOTAL BREECH EXTRACTION 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD 72.7 VACUUM EXTRACTION 72.71 VACUUM EXTRACTION WITH EPISIOTOMY 72.79 OTHER VACUUM EXTRACTION 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY 73.0 ARTIFICIAL RUPTURE OF MEMBRANES 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES 73.1 OTHER SURGICAL INDUCTION OF LABOR 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION 73.3 FAILED FORCEPS 73.4 MEDICAL INDUCTION OF LABOR 73.5 MANUALLY ASSISTED DELIVERY 73.51 MANUAL ROTATION OF FETAL HEAD 73.59 OTHER MANUALLY ASSISTED DELIVERY 73.6 EPISIOTOMY 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY 73.9 OTHER OPERATIONS ASSISTING DELIVERY 73.91 EXTERNAL VERSION ASSISTING DELIVERY 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD 73.93 INCISION OF CERVIX TO ASSIST DELIVERY 73.94 PUBIOTOMY TO ASSIST DELIVERY 73.99 OTHER OPERATIONS ASSISTING DELIVERY 74.0 CLASSICAL CESAREAN SECTION 74.1 LOW CERVICAL CESAREAN SECTION 74.2 EXTRAPERITONEAL CESAREAN SECTION 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE 75.4 MANUAL REMOVAL OF RETAINED PLACENTA 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM 75.9 OTHER OBSTETRIC OPERATIONS

Optum MarketScan

BEFORE PS MATCHING





The c-statistics for the propensity score model, pre-matching was 0.781.

The post-matching c-statistic was 0.578.

The c-statistics for the propensity score model, pre-matching was 0.758.

The post-matching c-statistic was 0.554.

AFTER PS MATCHING





| | | | | Uni | matched | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optu | n | | Markets | can | | POOLED | | |
| Variable | Risedronate | Teriparatide | St. Diff. | Risedronate | Teriparatide | St. Diff. | Risedronate | Teriparatide | St. Diff. |
| Number of patients | 3,875 | 853 | | 6,464 | 1,565 | | 10,339 | 2,418 | |
| Demographic characteristics | | | | | | | | | |
| Age | | | | | | | | | |
| mean (sd) | 72.33 (10.26) | 71.04 (10.08) | 0.127 | 70.65 (12.30) | 70.66 (11.23) | -0.001 | 71.28 (11.58) | 70.79 (10.84) | 0.044 |
| median [IQR] | 74.00 [65.00, 81.00] | 72.00 [63.00, 79.50] | 0.197 | 71.00 [60.00, 81.00] | 71.00 [62.00, 80.00] | 0.000 | 72.12 (11.58) | 71.35 (10.84) | 0.069 |
| Age categories | 46 (4. 20() | 42 (4 40() | 0.040 | 120 (2.10() | 24/4 50/1 | 0.045 | 404 (4.00() | 025 (4 50() | 0.024 |
| <50; n (%) | 46 (1.2%) | 12 (1.4%)<br>250 (29.3%) | -0.018<br>-0.134 | 138 (2.1%)<br>2,387 (36.9%) | 24 (1.5%) | 0.045<br>0.069 | 184 (1.8%)<br>3,293 (31.9%) | 036 (1.5%) | 0.024<br>-0.004 |
| 50 - 64; n (%)<br>65 - 79; n (%) | 906 (23.4%)<br>1,787 (46.1%) | 378 (44.3%) | 0.036 | 2,013 (31.1%) | 526 (33.6%)<br>616 (39.4%) | -0.174 | 3,800 (36.8%) | 776 (32.1%)<br>994 (41.1%) | -0.004 |
| >= 80; n (%) | 1,136 (29.3%) | 213 (25.0%) | 0.030 | 1,926 (29.8%) | 399 (25.5%) | 0.096 | 3,062 (29.6%) | 612 (25.3%) | 0.096 |
| Region | 1,130 (23.370) | 213 (23.070) | 0.037 | 1,520 (25.070) | 333 (23.370) | 0.050 | 3,002 (23.070) | 012 (23.370) | 0.050 |
| Northeast; n (%) | 352 (9.1%) | 78 (9.1%) | 0.000 | 1,422 (22.0%) | 260 (16.6%) | 0.137 | 1,774 (17.2%) | 338 (14.0%) | 0.088 |
| Midwest; n (%) | 580 (15.0%) | 149 (17.5%) | -0.068 | 1,712 (26.5%) | 475 (30.4%) | -0.087 | 2,292 (22.2%) | 624 (25.8%) | -0.084 |
| South; n (%) | 1,522 (39.3%) | 350 (41.0%) | -0.035 | 2,085 (32.3%) | 593 (37.9%) | -0.118 | 3,607 (34.9%) | 943 (39.0%) | -0.085 |
| West; n (%) | 1,421 (36.7%) | 276 (32.4%) | 0.091 | 1,245 (19.3%) | 237 (15.1%) | 0.111 | 2,666 (25.8%) | 513 (21.2%) | 0.109 |
| Calendar Time year of initiation | | | | | | | | | |
| Jan 2004 - Dec 2006; n (%) | 288 (7.4%) | 44 (5.2%) | 0.091 | 1,402 (21.7%) | 150 (9.6%) | 0.338 | 1,690 (16.3%) | 194 (8.0%) | 0.256 |
| Jan 2007 - Dec 2009; n (%) | 1,164 (30.0%) | 126 (14.8%) | 0.371 | 1,880 (29.1%) | 301 (19.2%) | 0.233 | 3,044 (29.4%) | 427 (17.7%) | 0.278 |
| Jan 2010 - Dec 2012; n (%) | 1,142 (29.5%) | 157 (18.4%) | 0.262 | 1,629 (25.2%) | 416 (26.6%) | -0.032 | 2,771 (26.8%) | 573 (23.7%) | 0.071 |
| Jan 2013 - Dec 2015; n (%) | 658 (17.0%) | 232 (27.2%) | -0.248 | 1,014 (15.7%) | 416 (26.6%) | -0.269 | 1,672 (16.2%) | 648 (26.8%) | -0.260 |
| Jan 2016 - Mar 2020; n (%) # | 623 (16.1%) | 294 (34.5%) | -0.433 | 539 (8.3%) | 282 (18.0%) | -0.027 | 1,162 (11.2%) | 576 (23.8%) | -0.336 |
| Race | | | | | | | | | |
| White; n (%) | 2,764 (71.3%) | 640 (75.0%) | -0.084 | NA | NA | NA | 2,764 (71.3%) | 640 (75.0%) | -0.084 |
| Black or African American; n (%) | 216 (5.6%) | 44 (5.2%) | 0.018 | NA | NA | NA | 216 (5.6%) | 44 (5.2%) | 0.018 |
| Asian; n (%) | 185 (4.8%) | 31 (3.6%) | 0.060<br>0.056 | NA<br>NA | NA<br>NA | NA<br>NA | 185 (4.8%) | 31 (3.6%) | 0.060<br>0.056 |
| Others; n (%) Metropolitan Statistical Area | 710 (18.3%) | 138 (16.2%) | 0.056 | NA | NA | NA | 710 (18.3%) | 138 (16.2%) | 0.056 |
| Urban; n (%) | NA | NA | NA | 4,979 (77.0%) | 1,173 (75.0%) | 0.047 | 4,979 (77.0%) | 1,173 (75.0%) | 0.047 |
| Rural; n (%) | NA<br>NA | NA<br>NA | NA | 37 (0.6%) | 41 (2.6%) | -0.160 | 37 (0.6%) | 41 (2.6%) | -0.160 |
| Unknown/Missing; n (%) | NA NA | NA | NA | 1,448 (22.4%) | 351 (22.4%) | 0.000 | 1,448 (22.4%) | 351 (22.4%) | 0.000 |
| General Health Related Measures | | 191 | | 1,110 (22.170) | 551 (22.170) | 0.000 | 1,110 (22.170) | 551 (22.170) | 0.000 |
| Smoking; n (%) | 355 (9.2%) | 123 (14.4%) | -0.162 | 290 (4.5%) | 108 (6.9%) | -0.104 | 645 (6.2%) | 231 (9.6%) | -0.126 |
| Obesity or Overweight; n (%) | 259 (6.7%) | 85 (10.0%) | -0.120 | 222 (3.4%) | 88 (5.6%) | -0.106 | 481 (4.7%) | 173 (7.2%) | -0.106 |
| Obesity; n (%) | 175 (4.5%) | 57 (6.7%) | -0.096 | 174 (2.7%) | 64 (4.1%) | -0.077 | 349 (3.4%) | 121 (5.0%) | -0.080 |
| Overweight; n (%) | 97 (2.5%) | 33 (3.9%) | -0.080 | 58 (0.9%) | 28 (1.8%) | -0.078 | 155 (1.5%) | 061 (2.5%) | -0.071 |
| Cardiovascular Measures | | | | | | | | | |
| Hypertension; n (%) | 2,391 (61.7%) | 503 (59.0%) | 0.055 | 2,945 (45.6%) | 744 (47.5%) | -0.038 | 5,336 (51.6%) | 1,247 (51.6%) | 0.000 |
| Hyperlipidemia; n (%) | 2,236 (57.7%) | 439 (51.5%) | 0.125 | 2,462 (38.1%) | 620 (39.6%) | -0.031 | 4,698 (45.4%) | 1,059 (43.8%) | 0.032 |
| Coronary artery disease (MI, angina, Coronary atherosclerosis and other forms of | 669 (17.3%) | 126 (14.8%) | 0.068 | 897 (13.9%) | 262 (16.7%) | -0.078 | 1,566 (15.1%) | 388 (16.0%) | -0.025 |
| chronic ischemic heart disease); n (%) | | | | | | | | | |
| Old MI; n (%) | 103 (2.7%) | 21 (2.5%) | 0.013 | 62 (1.0%) | 20 (1.3%) | -0.028 | 165 (1.6%) | 041 (1.7%) | -0.008 |
| Acute MI; n (%) | 48 (1.2%) | 6 (0.7%) | 0.052 | 65 (1.0%) | 18 (1.2%) | -0.019 | 113 (1.1%) | 024 (1.0%) | 0.010 |
| ACS/unstable angina; n (%) Stable angina; n (%) | 63 (1.6%) | 10 (1.2%) | 0.034<br>0.063 | 90 (1.4%)<br>145 (2.2%) | 25 (1.6%)<br>37 (2.4%) | -0.016<br>-0.013 | 153 (1.5%)<br>264 (2.6%) | 035 (1.4%)<br>055 (2.3%) | 0.008<br>0.019 |
| Coronary atherosclerosis and other CHD; n (%) | 119 (3.1%) | 18 (2.1%) | 0.003 | 800 (12.4%) | 232 (14.8%) | -0.013 | 1,376 (13.3%) | 339 (14.0%) | -0.020 |
| History of CABG or PTCA; n (%) | 576 (14.9%)<br>104 (2.7%) | 107 (12.5%)<br>19 (2.2%) | 0.070 | 57 (0.9%) | 24 (1.5%) | -0.055 | 161 (1.6%) | 043 (1.8%) | -0.020 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%) | 290 (7.5%) | 61 (7.2%) | 0.032 | 415 (6.4%) | 94 (6.0%) | 0.033 | 705 (6.8%) | 155 (6.4%) | 0.016 |
| Stroke (Ischemic or hemorrhagic); n (%) | 160 (4.1%) | 39 (4.6%) | -0.025 | 260 (4.0%) | 54 (3.5%) | 0.026 | 420 (4.1%) | 093 (3.8%) | 0.015 |
| TIA: n (%) | 126 (3.3%) | 20 (2.3%) | 0.061 | 187 (2.9%) | 47 (3.0%) | -0.006 | 313 (3.0%) | 067 (2.8%) | 0.012 |
| Late effects of cerebrovascular disease; n (%) | 95 (2.5%) | 27 (3.2%) | -0.042 | 92 (1.4%) | 20 (1.3%) | 0.009 | 187 (1.8%) | 047 (1.9%) | -0.007 |
| Heart Failure; n (%) | 279 (7.2%) | 44 (5.2%) | 0.083 | 466 (7.2%) | 128 (8.2%) | -0.038 | 745 (7.2%) | 172 (7.1%) | 0.004 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 310 (8.0%) | 73 (8.6%) | -0.022 | 393 (6.1%) | 102 (6.5%) | -0.016 | 703 (6.8%) | 175 (7.2%) | -0.016 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%) | 593 (15.3%) | 154 (18.1%) | -0.075 | 906 (14.0%) | 259 (16.5%) | -0.070 | 1,499 (14.5%) | 413 (17.1%) | -0.071 |
| Atrial fibrillation; n (%) | 323 (8.3%) | 81 (9.5%) | -0.042 | 492 (7.6%) | 153 (9.8%) | -0.078 | 815 (7.9%) | 234 (9.7%) | -0.064 |
| Other cardiac dysrhythmia; n (%) | 416 (10.7%) | 121 (14.2%) | -0.106 | 602 (9.3%) | 175 (11.2%) | -0.063 | 1,018 (9.8%) | 296 (12.2%) | -0.077 |
| Diabetes Related Measures | | | | | | | | | |
| Diabetes with or w/o complications; n (%) | 763 (19.7%) | 175 (20.5%) | -0.020 | 1,010 (15.6%) | 277 (17.7%) | -0.056 | 1,773 (17.1%) | 452 (18.7%) | -0.042 |
| Diabetes mellitus without mention of complications; n (%) | 689 (17.8%) | 151 (17.7%) | 0.003 | 891 (13.8%) | 236 (15.1%) | -0.037 | 1,580 (15.3%) | 387 (16.0%) | -0.019 |
| Diabetes with specified complications; n (%) | 248 (6.4%) | 61 (7.2%) | -0.032 | 292 (4.5%) | 101 (6.5%) | -0.088 | 540 (5.2%) | 162 (6.7%) | -0.063 |
| Diabetes with unspecified complications; n (%) | 34 (0.9%) | 6 (0.7%) | 0.022 | 41 (0.6%) | 14 (0.9%) | -0.035 | 075 (0.7%) | 020 (0.8%) | -0.012 |
| Hypoglycemia; n (%) GI Conditions | 54 (1.4%) | 17 (2.0%) | -0.046 | 56 (0.9%) | 24 (1.5%) | -0.055 | 110 (1.1%) | 041 (1.7%) | -0.051 |
| Upper GI (Diseases of esophagus, stomach and duodenum); n (%) | 852 (22.0%) | 254 (29.8%) | -0.179 | 861 (13.3%) | 334 (21.3%) | -0.213 | 1,713 (16.6%) | 588 (24.3%) | -0.192 |
| GI bleeding; n (%) | 167 (4.3%) | 30 (3.5%) | 0.041 | 269 (4.2%) | 54 (3.5%) | 0.036 | 436 (4.2%) | 084 (3.5%) | 0.036 |

| | 1 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Eating disorders, Non-infective enteritis and colitis, postoperative disorders of the digestive system; n (%) | 616 (15.9%) | 165 (19.3%) | -0.089 | 794 (12.3%) | 238 (15.2%) | -0.084 | 1,410 (13.6%) | 403 (16.7%) | -0.087 |
| Eating disorders (Anorexia and Bulimia); n (%) | 238 (6.1%) | 68 (8.0%) | -0.074 | 190 (2.9%) | 74 (4.7%) | -0.094 | 428 (4.1%) | 142 (5.9%) | -0.083 |
| Non-infective enteritis and colitis; n (%) | 323 (8.3%) | 85 (10.0%) | -0.059 | 469 (7.3%) | 143 (9.1%) | -0.066 | 792 (7.7%) | 228 (9.4%) | -0.061 |
| Intraoperative and postprocedural complications and disorders of digestive system; | 158 (4.1%) | 38 (4.5%) | -0.020 | 257 (4.0%) | 55 (3.5%) | 0.026 | 415 (4.0%) | 093 (3.8%) | 0.010 |
| n (%) Disorders of gallbladder, biliary tract and pancreas; n (%) | 100 (2.6%) | 40 (4.7%) | -0.112 | 188 (2.9%) | 57 (3.6%) | -0.039 | 288 (2.8%) | 097 (4.0%) | -0.066 |
| Rheumatic Conditions | 100 (2.0%) | 40 (4.776) | -0.112 | 100 (2.5%) | 37 (3.0%) | -0.033 | 200 (2.070) | 037 (4.078) | -0.000 |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n (%) | 317 (8.2%) | 116 (13.6%) | -0.174 | 426 (6.6%) | 184 (11.8%) | -0.181 | 743 (7.2%) | 300 (12.4%) | -0.176 |
| Osteoarthrosis; n (%) | 1,276 (32.9%) | 347 (40.7%) | -0.162 | 1,580 (24.4%) | 528 (33.7%) | -0.206 | 2,856 (27.6%) | 875 (36.2%) | -0.185 |
| Other rheumatic disorders (including gout); n (%) | 2,635 (68.0%) | 630 (73.9%) | -0.130 | 4,107 (63.5%) | 1,129 (72.1%) | -0.185 | 6,742 (65.2%) | 1,759 (72.7%) | -0.163 |
| Gout and other crystal arthropathies; n (%) | 80 (2.1%) | 15 (1.8%) | 0.022 | 68 (1.1%) | 29 (1.9%) | -0.066 | 148 (1.4%) | 044 (1.8%) | -0.032 |
| Other rheumatic disorders; n (%) | 2,620 (67.6%) | 628 (73.6%) | -0.132 | 4,090 (63.3%) | 1,123 (71.8%) | -0.182 | 6,710 (64.9%) | 1,751 (72.4%) | -0.162 |
| Neuro Conditions Parkinson's disease; n (%) | 10 (0.3%) | 1 (0.1%) | 0.045 | 8 (0.1%) | 2 (0.1%) | 0.000 | 018 (0.2%) | 003 (0.1%) | 0.026 |
| Alzheimer and other Dementia Disease ; n (%) | 373 (9.6%) | 62 (7.3%) | 0.043 | 462 (7.1%) | 100 (6.4%) | 0.000 | 835 (8.1%) | 162 (6.7%) | 0.026 |
| Seizure disorders (epilepsy); n (%) | 61 (1.6%) | 21 (2.5%) | -0.064 | 73 (1.1%) | 31 (2.0%) | -0.073 | 134 (1.3%) | 052 (2.2%) | -0.069 |
| Delirium/Psychosis; n (%) | 148 (3.8%) | 33 (3.9%) | -0.005 | 192 (3.0%) | 62 (4.0%) | -0.054 | 340 (3.3%) | 095 (3.9%) | -0.032 |
| Other Conditions | | | | | | | | | |
| Vitamin D deficiency; n (%) | 633 (16.3%) | 250 (29.3%) | -0.314 | 546 (8.4%) | 263 (16.8%) | -0.255 | 1,179 (11.4%) | 513 (21.2%) | -0.268 |
| Liver disease; n (%) | 128 (3.3%) | 37 (4.3%) | -0.052 | 194 (3.0%) | 56 (3.6%) | -0.034 | 322 (3.1%) | 093 (3.8%) | -0.038 |
| Chronic kidney disease stages I-III; n (%) | 414 (10.7%) | 81 (9.5%) | 0.040 | 181 (2.8%) | 72 (4.6%) | -0.095 | 595 (5.8%) | 153 (6.3%) | -0.021 |
| Chronic kidney disease stages IV-V, ESRD; n (%) Premature menopause; n (%) | 130 (3.4%)<br>5 (0.1%) | 18 (2.1%)<br>3 (0.4%) | 0.080<br>-0.060 | 60 (0.9%)<br>9 (0.1%) | 27 (1.7%)<br>1 (0.1%) | -0.071<br>0.000 | 190 (1.8%)<br>014 (0.1%) | 045 (1.9%)<br>004 (0.2%) | -0.007<br>-0.026 |
| Oophorectomy; n (%) | 5 (0.1%) | 0 (0.0%) | 0.045 | 1 (0.0%) | 1 (0.1%) | -0.045 | 006 (0.1%) | 004 (0.2%) | 0.026 |
| COPD; n (%) | 623 (16.1%) | 142 (16.6%) | -0.014 | 798 (12.3%) | 244 (15.6%) | -0.095 | 1,421 (13.7%) | 386 (16.0%) | -0.065 |
| Asthma; n (%) | 384 (9.9%) | 102 (12.0%) | -0.067 | 484 (7.5%) | 147 (9.4%) | -0.068 | 868 (8.4%) | 249 (10.3%) | -0.065 |
| Obstructive sleep apnea; n (%) | 151 (3.9%) | 60 (7.0%) | -0.137 | 143 (2.2%) | 62 (4.0%) | -0.104 | 294 (2.8%) | 122 (5.0%) | -0.114 |
| Syncope; n (%) | 215 (5.5%) | 49 (5.7%) | -0.009 | 343 (5.3%) | 89 (5.7%) | -0.018 | 558 (5.4%) | 138 (5.7%) | -0.013 |
| Falls; n (%) | 499 (12.9%) | 180 (21.1%) | -0.220 | 173 (2.7%) | 128 (8.2%) | -0.244 | 672 (6.5%) | 308 (12.7%) | -0.212 |
| VTE; n (%) | 142 (3.7%) | 36 (4.2%) | -0.026 | 203 (3.1%) | 58 (3.7%) | -0.033 | 345 (3.3%) | 094 (3.9%) | -0.032 |
| Gait abnormality; n (%) | 498 (12.9%)<br>1,260 (32.5%) | 179 (21.0%)<br>279 (32.7%) | -0.217<br>-0.004 | 578 (8.9%)<br>1,720 (26.6%) | 202 (12.9%)<br>344 (22.0%) | -0.129<br>0.107 | 1,076 (10.4%)<br>2,980 (28.8%) | 381 (15.8%)<br>623 (25.8%) | -0.161<br>0.067 |
| Osteopenia; n (%) History of hip and femur fractures; n (%) | 1,260 (32.5%) | 279 (32.7%)<br>66 (7.7%) | -0.004 | 280 (4.3%) | 344 (22.0%)<br>141 (9.0%) | -0.189 | 2,980 (28.8%)<br>442 (4.3%) | 207 (8.6%) | -0.176 |
| Other Fractures ; n (%) | 267 (6.9%) | 123 (14.4%) | -0.245 | 425 (6.6%) | 199 (12.7%) | -0.208 | 692 (6.7%) | 322 (13.3%) | -0.221 |
| Glucocorticoid-Induced Osteoporosis; n (%) | 4 (0.1%) | 3 (0.4%) | -0.060 | 1 (0.0%) | 2 (0.1%) | -0.045 | 005 (0.0%) | 005 (0.2%) | -0.063 |
| Combined comorbidity score | | | | | | | | | |
| mean (sd) | 1.03 (2.10) | 1.28 (2.22) | -0.116 | 0.66 (1.57) | 0.92 (1.78) | -0.155 | 0.80 (1.79) | 1.05 (1.95) | -0.134 |
| median [IQR] | 0.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | -0.463 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.00 (1.79) | 0.35 (1.95) | -0.187 |
| Frailty Score: Empirical Version 365 days as Categories | 4 500 (44 20/) | 272 (42 69/) | 0.047 | 2 520 (40 70) | 507 (22 40() | 0.472 | 4 220 (40 00() | 070 (25 40() | 0.000 |
| <0.12908; n (%)<br>0.12908 - 0.1631167; n (%) | 1,600 (41.3%)<br>852 (22.0%) | 372 (43.6%)<br>173 (20.3%) | -0.047<br>0.042 | 2,630 (40.7%)<br>1,510 (23.4%) | 507 (32.4%)<br>342 (21.9%) | 0.173<br>0.036 | 4,230 (40.9%)<br>2,362 (22.8%) | 879 (36.4%)<br>515 (21.3%) | 0.093<br>0.036 |
| >=0.1631167; n (%) | 1,423 (36.7%) | 308 (36.1%) | 0.012 | 2,324 (36.0%) | 716 (45.8%) | -0.200 | 3,747 (36.2%) | 1,024 (42.3%) | -0.125 |
| Medication Use | -, (, | () | | _,== : (==:=,=, | . == ( , | | o, (o o · = · - ) | _,==:(:=:=,-, | |
| Use of oral corticosteroids; n (%) | 1,089 (28.1%) | 314 (36.8%) | -0.187 | 1,859 (28.8%) | 572 (36.5%) | -0.165 | 2,948 (28.5%) | 886 (36.6%) | -0.174 |
| Use of antidepressants; n (%) | 1,247 (32.2%) | 327 (38.3%) | -0.128 | 2,143 (33.2%) | 654 (41.8%) | -0.178 | 3,390 (32.8%) | 981 (40.6%) | -0.162 |
| Use of anticonvulsants; n (%) | 565 (14.6%) | 180 (21.1%) | -0.170 | 904 (14.0%) | 376 (24.0%) | -0.257 | 1,469 (14.2%) | 556 (23.0%) | -0.228 |
| Use of beta blocker OR calcium channel blocker; n (%) | 1,270 (32.8%) | 270 (31.7%) | 0.024 | 2,060 (31.9%) | 537 (34.3%) | -0.051 | 3,330 (32.2%) | 807 (33.4%) | -0.026 |
| Use of PPIs; n (%) Use of opioids; n (%) | 965 (24.9%)<br>1,674 (43.2%) | 254 (29.8%)<br>488 (57.2%) | -0.110<br>-0.283 | 1,761 (27.2%)<br>2,972 (46.0%) | 569 (36.4%)<br>976 (62.4%) | -0.199<br>-0.334 | 2,726 (26.4%)<br>4,646 (44.9%) | 823 (34.0%)<br>1,464 (60.5%) | -0.166<br>-0.316 |
| Use of antipsychotics; n (%) | 108 (2.8%) | 28 (3.3%) | -0.029 | 230 (3.6%) | 61 (3.9%) | -0.016 | 338 (3.3%) | 089 (3.7%) | -0.022 |
| Use of anxiolytics/hypnotics; n (%) | 435 (11.2%) | 91 (10.7%) | 0.016 | 816 (12.6%) | 255 (16.3%) | -0.105 | 1,251 (12.1%) | 346 (14.3%) | -0.065 |
| Use of dementia meds; n (%) | 219 (5.7%) | 34 (4.0%) | 0.079 | 349 (5.4%) | 77 (4.9%) | 0.023 | 568 (5.5%) | 111 (4.6%) | 0.041 |
| Use of antiparkinsonian meds; n (%) | 127 (3.3%) | 33 (3.9%) | -0.032 | 226 (3.5%) | 67 (4.3%) | -0.041 | 353 (3.4%) | 100 (4.1%) | -0.037 |
| Use of Benzodiazepine; n (%) | 568 (14.7%) | 200 (23.4%) | -0.223 | 1,491 (23.1%) | 433 (27.7%) | -0.106 | 2,059 (19.9%) | 633 (26.2%) | -0.150 |
| All antidiabetic medications; n (%) | 439 (11.3%) | 82 (9.6%) | 0.056 | 670 (10.4%) | 188 (12.0%) | -0.051 | 1,109 (10.7%) | 270 (11.2%) | -0.016 |
| ACEI/ARB; n (%) | 1,555 (40.1%) | 280 (32.8%) | 0.152 | 2,234 (34.6%) | 527 (33.7%) | 0.019 | 3,789 (36.6%) | 807 (33.4%) | 0.067 |
| Use of Anticoagulants; n (%) Use of Amiodarone; n (%) | 301 (7.8%)<br>36 (0.9%) | 81 (9.5%)<br>10 (1.2%) | -0.061<br>-0.029 | 548 (8.5%)<br>81 (1.3%) | 176 (11.2%)<br>26 (1.7%) | -0.091<br>-0.033 | 849 (8.2%)<br>117 (1.1%) | 257 (10.6%)<br>036 (1.5%) | -0.082<br>-0.035 |
| Digoxin; n (%) | 92 (2.4%) | 17 (2.0%) | 0.029 | 233 (3.6%) | 45 (2.9%) | 0.039 | 325 (3.1%) | 062 (2.6%) | 0.030 |
| Use of Diuretics; n (%) | 1,273 (32.9%) | 251 (29.4%) | 0.076 | 2,096 (32.4%) | 515 (32.9%) | -0.011 | 3,369 (32.6%) | 766 (31.7%) | 0.019 |
| Use of Aspirin; n (%) | 24 (0.6%) | 6 (0.7%) | -0.012 | 90 (1.4%) | 25 (1.6%) | -0.016 | 114 (1.1%) | 031 (1.3%) | -0.018 |
| NSAIDs (NOT including aspirin); n (%) | 807 (20.8%) | 218 (25.6%) | -0.114 | 1,496 (23.1%) | 365 (23.3%) | -0.005 | 2,303 (22.3%) | 583 (24.1%) | -0.043 |
| HRT (Use of estrogens, progestins, androgens); n (%) | 240 (6.2%) | 50 (5.9%) | 0.013 | 445 (6.9%) | 102 (6.5%) | 0.016 | 685 (6.6%) | 152 (6.3%) | 0.012 |
| Other Pressors; n (%) | 24 (0.6%) | 5 (0.6%) | 0.000 | 38 (0.6%) | 24 (1.5%) | -0.088 | 062 (0.6%) | 029 (1.2%) | -0.064 |
| Use of Statins; n (%) | 1,599 (41.3%) | 276 (32.4%) | 0.185 | 2,393 (37.0%) | 568 (36.3%) | 0.015<br>-0.034 | 3,992 (38.6%) | 844 (34.9%) | 0.077<br>-0.042 |
| Selective Estrogen Receptor Modulators (SERMs); n (%) | 61 (1.6%) | 19 (2.2%) | -0.044 | 128 (2.0%) | 39 (2.5%) | -0.034 | 189 (1.8%) | 058 (2.4%) | -0.042 |

| In the second second | ī | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Healthcare Utilization Measures | | | | | | | | | |
| Use of any drugs claims | | | | | | | | | |
| mean (sd) | 21.89 (16.94) | 25.76 (18.99) | -0.215 | 20.60 (16.91) | 26.58 (19.21) | -0.330 | 21.08 (16.92) | 26.29 (19.13) | -0.289 |
| Number of office visits | | | | | | | | | |
| mean (sd) | 8.64 (6.54) | 12.05 (7.91) | -0.470 | 9.37 (7.10) | 12.43 (8.14) | -0.401 | 9.10 (6.90) | 12.30 (8.06) | -0.427 |
| Number of ED visits | | | | | | | | | |
| mean (sd) | 0.59 (1.17) | 0.77 (1.14) | -0.156 | 0.49 (1.14) | 0.65 (1.25) | -0.134 | 0.53 (1.15) | 0.69 (1.21) | -0.136 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 0.32 (0.86) | 0.48 (1.01) | -0.171 | 1.83 (6.41) | 2.30 (5.88) | -0.076 | 1.26 (5.10) | 1.66 (4.77) | -0.081 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 55 (1.4%) | 21 (2.5%) | -0.080 | 125 (1.9%) | 37 (2.4%) | -0.034 | 180 (1.7%) | 058 (2.4%) | -0.049 |
| Old hospitalizations (-450 to -31 days); n (%) | 579 (14.9%) | 200 (23.4%) | -0.217 | 1,301 (20.1%) | 420 (26.8%) | -0.159 | 1,880 (18.2%) | 620 (25.6%) | -0.180 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.14 (0.67) | 0.52 (1.28) | -0.372 | 1.52 (2.62) | 1.77 (2.97) | -0.089 | 1.00 (2.11) | 1.33 (2.51) | -0.142 |
| Number of DXA test performed | | | | | | | | | |
| mean (sd) | 0.57 (0.57) | 0.74 (0.56) | -0.301 | 0.41 (0.51) | 0.50 (0.53) | -0.173 | 0.47 (0.53) | 0.58 (0.54) | -0.206 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 3.68 (14.88) | 5.21 (17.30) | -0.095 | 1.83 (6.41) | 2.30 (5.88) | -0.076 | 2.52 (10.42) | 3.33 (11.31) | -0.074 |
| Occurrence of basic or comprehensive blood chemistry test; n (%) | 2,611 (67.4%) | 660 (77.4%) | -0.012 | 2,508 (38.8%) | 720 (46.0%) | -0.146 | 5,119 (49.5%) | 1,380 (57.1%) | -0.153 |
| Number of HbA1C test ordered | | | | | | | | | |
| mean (sd) | 0.55 (1.14) | 0.53 (1.13) | 0.018 | 0.28 (0.84) | 0.27 (0.79) | 0.012 | 0.38 (0.96) | 0.36 (0.92) | 0.021 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) | 305 (7.9%) | 77 (9.0%) | -0.040 | 649 (10.0%) | 146 (9.3%) | 0.024 | 954 (9.2%) | 223 (9.2%) | 0.000 |
| Number of Mammograms (Breast cancer screening); n (%) | 1,955 (50.5%) | 408 (47.8%) | 0.054 | 3,028 (46.8%) | 583 (37.3%) | 0.193 | 4,983 (48.2%) | 991 (41.0%) | 0.145 |
| Number of Pap smear (Cervical cancer screening); n (%) | 873 (22.5%) | 153 (17.9%) | 0.115 | 1,683 (26.0%) | 279 (17.8%) | 0.199 | 2,556 (24.7%) | 432 (17.9%) | 0.167 |
| Flu vaccine; n (%) | 1,331 (34.3%) | 318 (37.3%) | -0.063 | 1,329 (20.6%) | 349 (22.3%) | -0.041 | 2,660 (25.7%) | 667 (27.6%) | -0.043 |
| Pneumococcal vaccine; n (%) | 493 (12.7%) | 168 (19.7%) | -0.191 | 417 (6.5%) | 155 (9.9%) | -0.124 | 910 (8.8%) | 323 (13.4%) | -0.147 |
| Copay for pharmacy cost (charges in U.S. \$) | | | | | | | | | |
| mean (sd) | 32.47 (33.44) | 39.58 (80.44) | -0.115 | 24.71 (28.10) | 21.31 (23.34) | 0.132 | 27.62 (30.21) | 27.76 (51.33) | -0.003 |
| median [IQR] | 24.33 [13.75, 40.90] | 25.00 [12.09, 41.51] | -0.011 | 18.73 [8.26, 32.00] | 16.84 [7.92, 28.17] | 0.073 | 20.83 (30.21) | 19.72 (51.33) | 0.026 |
| Missing; n (%) | 0 (0.0%) | 1 (0.1%) | -0.018 | 0 (0.0%) | 5 (0.3%) | -0.078 | 000 (0.0%) | 006 (0.2%) | -0.063 |
| Business Type | , , | . , | | , , | , , | | , , | , , | |
| Commercial; n (%) | 1,313 (33.9%) | 344 (40.3%) | -0.133 | NA | NA | NA | 1,313 (33.9%) | 344 (40.3%) | -0.133 |
| Medicare; n (%) | 2,562 (66.1%) | 509 (59.7%) | 0.133 | NA | NA | NA | 2,562 (66.1%) | 509 (59.7%) | 0.133 |
| Insurance Plan Type | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ( , | | | | | , ( , | , | |
| Comprehensive; n (%) | NA | NA | NA | 1,771 (27.4%) | 476 (30.4%) | -0.066 | 1,771 (27.4%) | 476 (30.4%) | -0.066 |
| HMO; n (%) | NA | NA | NA | 922 (14.3%) | 109 (7.0%) | 0.238 | 922 (14.3%) | 109 (7.0%) | 0.238 |
| PPO; n (%) | NA NA | NA NA | NA | 3,087 (47.8%) | 780 (49.8%) | -0.040 | 3,087 (47.8%) | 780 (49.8%) | -0.040 |
| Others; n (%) | NA NA | NA<br>NA | NA<br>NA | 684 (10.6%) | 200 (12.8%) | -0.068 | 684 (10.6%) | 200 (12.8%) | -0.068 |
| | I INA | .40 | .4/5 | 33.(10.070) | 200 (12.070) | 5.500 | 33.(10.070) | 200 (12.070) | 0.000 |

Aetion link to Optum results: https://bwh-dope.aetion.com/projects/details/1640/rwrs/67726
Aetion link to Marketscan results: https://bwh-dope.aetion.com/projects/details/1641/rwrs/67727

#The last cohort entry date in Optum is Mar 31, 2020 and in Marketscan is Dec 31, 2018

| | | PS-matched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Or | otum | Circu | Marke | | POC | OLED | | |
| Variable | Risedronate | Teriparatide | St. Diff. | Risedronate | Teriparatide | St. Diff. | Risedronate | Teriparatide | St. Diff. |
| Number of patients | 74 | 7 747 | | 1,420 | 1,420 | | 2,167 | 2,167 | |
| Demographic characteristics | | | | | | | | | |
| Age | | | | | | | | | |
| mean (sd) | 71.16 (10.45) | 71.32 (10.12) | -0.016 | 70.57 (11.42) | 70.82 (11.22) | -0.022 | 70.77 (11.10) | 70.99 (10.85) | -0.020 |
| median [IQR] | 73.00 [63.00, 79.00] | 72.00 [63.00, 80.00] | 0.097 | 71.00 [61.00, 79.00] | 71.00 [62.00, 80.00] | 0.000 | 71.69 (11.10) | 71.34 (10.85) | 0.032 |
| Age categories* | | | | | | | | | |
| <50; n (%) | 8 (1.1%) | 12 (1.6%) | -0.043 | 22 (1.5%) | 23 (1.6%) | -0.008 | 030 (1.4%) | 035 (1.6%) | -0.016 |
| 50 - 64; n (%) | 207 (27.7%) | 208 (27.8%) | -0.002 | 478 (33.7%) | 472 (33.2%) | 0.011 | 685 (31.6%) | 680 (31.4%) | 0.004 |
| 65 - 79; n (%) | 350 (46.9%) | 333 (44.6%) | 0.046 | 571 (40.2%) | 551 (38.8%) | 0.029 | 921 (42.5%) | 884 (40.8%) | 0.034 |
| >= 80; n (%) | 182 (24.4%) | 194 (26.0%) | -0.037 | 349 (24.6%) | 374 (26.3%) | -0.039 | 531 (24.5%) | 568 (26.2%) | -0.039 |
| Region* | | | | | | | | | |
| Northeast; n (%) | 73 (9.8%) | 69 (9.2%) | 0.020 | 267 (18.8%) | 250 (17.6%) | 0.031 | 340 (15.7%) | 319 (14.7%) | 0.028 |
| Midwest; n (%) | 117 (15.7%) | 125 (16.7%) | -0.027 | 402 (28.3%) | 419 (29.5%) | -0.026 | 519 (24.0%) | 544 (25.1%) | -0.026 |
| South; n (%) | 317 (42.4%) | 302 (40.4%) | 0.041 | 545 (38.4%) | 530 (37.3%) | 0.023 | 862 (39.8%) | 832 (38.4%) | 0.029 |
| West; n (%) | 240 (32.1%) | 251 (33.6%) | -0.032 | 206 (14.5%) | 221 (15.6%) | -0.031 | 446 (20.6%) | 472 (21.8%) | -0.029 |
| Calendar Time year of initiation* | | 40 /= | 0.55 | 450/45 500 | 440/45 | | 40.47 | 100 (0) | |
| Jan 2004 - Dec 2006; n (%) | 44 (5.9%) | 43 (5.8%) | 0.004 | 150 (10.6%) | 149 (10.5%) | 0.003 | 194 (9.0%) | 192 (8.9%) | 0.004 |
| Jan 2007 - Dec 2009; n (%) | 122 (16.3%) | 123 (16.5%) | -0.005 | 297 (20.9%) | 292 (20.6%) | 0.007 | 419 (19.3%) | 415 (19.2%) | 0.003 |
| Jan 2010 - Dec 2012; n (%) | 158 (21.2%) | 153 (20.5%) | 0.017 | 402 (28.3%) | 397 (28.0%) | 0.007 | 560 (25.8%) | 550 (25.4%) | 0.009 |
| Jan 2013 - Dec 2015; n (%) | 190 (25.4%) | 200 (26.8%) | -0.032 | 369 (26.0%) | 361 (25.4%) | 0.014 | 559 (25.8%) | 561 (25.9%) | -0.002 |
| Jan 2016 - Mar 2020; n (%) # | 233 (31.2%) | 228 (30.5%) | 0.015 | 202 (14.2%) | 221 (15.6%) | -0.039 | 435 (20.1%) | 449 (20.7%) | -0.015 |
| Race* | | | | | | | | | |
| White; n (%) | 562 (75.2%) | 556 (74.4%) | 0.018 | NA | NA | NA | 562 (75.2%) | 556 (74.4%) | 0.018 |
| Black or African American; n (%) | 43 (5.8%) | 40 (5.4%) | 0.017 | NA | NA | NA | 43 (5.8%) | 40 (5.4%) | 0.017 |
| Asian; n (%) | 29 (3.9%) | 30 (4.0%) | -0.005 | NA | NA | NA | 29 (3.9%) | 30 (4.0%) | -0.005 |
| Others; n (%) | 113 (15.1%) | 121 (16.2%) | -0.030 | NA | NA | NA | 113 (15.1%) | 121 (16.2%) | -0.030 |
| Metropolitan Statistical Area* | | | | 4 000 (75 70) | 4 050 (75 00/) | | 4 000 (75 70) | 4 050 (75 00/) | |
| Urban; n (%) | NA<br>NA | NA | NA | 1,089 (76.7%) | 1,069 (75.3%) | 0.033 | 1,089 (76.7%) | 1,069 (75.3%) | 0.033 |
| Rural; n (%) | NA<br>NA | NA<br>NA | NA | 25 (1.8%) | 28 (2.0%) | -0.015 | 25 (1.8%) | 28 (2.0%) | -0.015 |
| Unknown/Missing; n (%) | INA | NA | NA | 306 (21.5%) | 323 (22.7%) | -0.029 | 306 (21.5%) | 323 (22.7%) | -0.029 |
| General Health Related Measures Smoking; n (%)* | 100 (13.4%) | 93 (12.4%) | 0.030 | 82 (5.8%) | 91 (6.4%) | -0.025 | 182 (8.4%) | 184 (8.5%) | -0.004 |
| | 61 (8.2%) | 68 (9.1%) | -0.032 | 68 (4.8%) | 76 (5.4%) | -0.023 | 129 (6.0%) | 144 (6.6%) | -0.004 |
| Obesity or Overweight; n (%)* | 44 (5.9%) | 45 (6.0%) | -0.032 | 51 (3.6%) | 76 (3.4%)<br>54 (3.8%) | -0.027 | 095 (4.4%) | 099 (4.6%) | -0.025 |
| Obesity; n (%) Overweight; n (%) | 22 (2.9%) | 27 (3.6%) | -0.004 | 22 (1.5%) | 26 (1.8%) | -0.011 | 044 (2.0%) | 053 (2.4%) | -0.010 |
| Cardiovascular Measures | 22 (2.370) | 27 (3.070) | -0.033 | 22 (1.370) | 20 (1.670) | -0.024 | 044 (2.078) | 055 (2.470) | -0.027 |
| Hypertension; n (%)* | 452 (60.5%) | 446 (59.7%) | 0.016 | 636 (44.8%) | 663 (46.7%) | -0.038 | 1,088 (50.2%) | 1,109 (51.2%) | -0.020 |
| Hyperlipidemia; n (%)* | 413 (55.3%) | 403 (53.9%) | 0.018 | 544 (38.3%) | 551 (38.8%) | -0.038 | 957 (44.2%) | 954 (44.0%) | 0.004 |
| Coronary artery disease (MI, angina, Coronary atherosclerosis and other forms of chronic | | | | | | | | | |
| ischemic heart disease); n (%)* | 117 (15.7%) | 111 (14.9%) | 0.022 | 212 (14.9%) | 222 (15.6%) | -0.019 | 329 (15.2%) | 333 (15.4%) | -0.006 |
| Old MI; n (%) | 14 (1.9%) | 20 (2.7%) | -0.053 | 18 (1.3%) | 17 (1.2%) | 0.009 | 032 (1.5%) | 037 (1.7%) | -0.016 |
| Acute MI; n (%) | 7 (0.9%) | 6 (0.8%) | 0.011 | 16 (1.1%) | 15 (1.1%) | 0.000 | 023 (1.1%) | 021 (1.0%) | 0.010 |
| ACS/unstable angina; n (%) | 12 (1.6%) | 9 (1.2%) | 0.034 | 16 (1.1%) | 23 (1.6%) | -0.043 | 028 (1.3%) | 032 (1.5%) | -0.017 |
| Stable angina; n (%) | 24 (3.2%) | 14 (1.9%) | 0.083 | 33 (2.3%) | 32 (2.3%) | 0.000 | 057 (2.6%) | 046 (2.1%) | 0.033 |
| Coronary atherosclerosis and other CHD; n (%) | 103 (13.8%) | 94 (12.6%) | 0.035 | 190 (13.4%) | 195 (13.7%) | -0.009 | 293 (13.5%) | 289 (13.3%) | 0.006 |
| History of CABG or PTCA; n (%) | 17 (2.3%) | 16 (2.1%) | 0.014 | 12 (0.8%) | 18 (1.3%) | -0.049 | 029 (1.3%) | 034 (1.6%) | -0.025 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%)* | 39 (5.2%) | 56 (7.5%) | -0.094 | 79 (5.6%) | 88 (6.2%) | -0.025 | 118 (5.4%) | 144 (6.6%) | -0.051 |
| Stroke (Ischemic or hemorrhagic); n (%) | 23 (3.1%) | 36 (4.8%) | -0.087 | 48 (3.4%) | 50 (3.5%) | -0.005 | 071 (3.3%) | 086 (4.0%) | -0.037 |
| TIA; n (%) | 19 (2.5%) | 18 (2.4%) | 0.006 | 36 (2.5%) | 45 (3.2%) | -0.042 | 055 (2.5%) | 063 (2.9%) | -0.025 |
| Late effects of cerebrovascular disease; n (%) | 12 (1.6%) | 24 (3.2%) | -0.105 | 17 (1.2%) | 19 (1.3%) | -0.009 | 029 (1.3%) | 043 (2.0%) | -0.055 |
| Heart Failure; n (%)* | 36 (4.8%) | 41 (5.5%) | -0.032 | 99 (7.0%) | 115 (8.1%) | -0.042 | 135 (6.2%) | 156 (7.2%) | -0.040 |
| Peripheral Vascular Disease (PVD) or PVD Surgery; n (%)* | 64 (8.6%) | 62 (8.3%) | 0.011 | 98 (6.9%) | 88 (6.2%) | 0.028 | 162 (7.5%) | 150 (6.9%) | 0.023 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%)* | 138 (18.5%) | 132 (17.7%) | 0.021 | 237 (16.7%) | 226 (15.9%) | 0.022 | 375 (17.3%) | 358 (16.5%) | 0.021 |
| Atrial fibrillation; n (%) | 76 (10.2%) | 70 (9.4%) | 0.027 | 128 (9.0%) | 131 (9.2%) | -0.007 | 204 (9.4%) | 201 (9.3%) | 0.003 |
| Other cardiac dysrhythmia; n (%) | 111 (14.9%) | 101 (13.5%) | 0.040 | 164 (11.5%) | 152 (10.7%) | 0.025 | 275 (12.7%) | 253 (11.7%) | 0.031 |
| Diabetes Related Measures | | | | | | | . , | | |
| Diabetes with or w/o complications; n (%)* | 161 (21.6%) | 149 (19.9%) | 0.042 | 255 (18.0%) | 240 (16.9%) | 0.029 | 416 (19.2%) | 389 (18.0%) | 0.031 |
| Diabetes mellitus without mention of complications; n (%) | 143 (19.1%) | 133 (17.8%) | 0.034 | 220 (15.5%) | 206 (14.5%) | 0.028 | 363 (16.8%) | 339 (15.6%) | 0.033 |
| Diabetes with specified complications; n (%) | 59 (7.9%) | 48 (6.4%) | 0.058 | 89 (6.3%) | 86 (6.1%) | 0.008 | 148 (6.8%) | 134 (6.2%) | 0.024 |
| Diabetes with unspecified complications; n (%) | 7 (0.9%) | 5 (0.7%) | 0.022 | 11 (0.8%) | 11 (0.8%) | 0.000 | 018 (0.8%) | 016 (0.7%) | 0.012 |

| Hypoglycemia; n (%)* | 9 (1.2%) | 15 (2.0%) | -0.064 | 17 (1.2%) | 22 (1.5%) | -0.026 | 026 (1.2%) | 037 (1.7%) | -0.042 |
|---|---|---|---|---|---|---|---|---|---|
| GI Conditions | | | | | | | | | |
| Upper GI (Diseases of esophagus, stomach and duodenum); n (%)* | 211 (28.2%) | 217 (29.0%) | -0.018 | 269 (18.9%) | 275 (19.4%) | -0.013 | 480 (22.2%) | 492 (22.7%) | -0.012 |
| GI bleeding; n (%)* | 26 (3.5%) | 27 (3.6%) | -0.005 | 58 (4.1%) | 51 (3.6%) | 0.026 | 084 (3.9%) | 078 (3.6%) | 0.016 |
| Eating disorders, Non-infective enteritis and colitis, postoperative disorders of the | 4.45 (4.0, 40() | 4.45 (40.50() | 0.002 | 205 (4.4.50() | 202 (4.4.20() | 0.006 | 254 (46 20() | 240 (45 40() | 0.002 |
| digestive system; n (%)* | 145 (19.4%) | 146 (19.5%) | -0.003 | 206 (14.5%) | 203 (14.3%) | 0.006 | 351 (16.2%) | 349 (16.1%) | 0.003 |
| Eating disorders (Anorexia and Bulimia); n (%) | 63 (8.4%) | 60 (8.0%) | 0.015 | 50 (3.5%) | 62 (4.4%) | -0.046 | 113 (5.2%) | 122 (5.6%) | -0.018 |
| Non-infective enteritis and colitis; n (%) | 69 (9.2%) | 75 (10.0%) | -0.027 | 133 (9.4%) | 124 (8.7%) | 0.024 | 202 (9.3%) | 199 (9.2%) | 0.003 |
| Intraoperative and postprocedural complications and disorders of digestive system; n | | | | | | 0.048 | | | |
| (%) | 34 (4.6%) | 34 (4.6%) | 0.000 | 58 (4.1%) | 46 (3.2%) | | 092 (4.2%) | 080 (3.7%) | 0.026 |
| Disorders of gallbladder, biliary tract and pancreas; n (%)* | 33 (4.4%) | 35 (4.7%) | -0.014 | 57 (4.0%) | 52 (3.7%) | 0.016 | 090 (4.2%) | 087 (4.0%) | 0.010 |
| Rheumatic Conditions | 55 (,,, | ( , -, | | (, | 0= (0, | | , | (, | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n (%)* | 95 (12.7%) | 97 (13.0%) | -0.009 | 163 (11.5%) | 150 (10.6%) | 0.029 | 258 (11.9%) | 247 (11.4%) | 0.016 |
| Osteoarthrosis; n (%)* | 283 (37.9%) | 298 (39.9%) | -0.041 | 445 (31.3%) | 456 (32.1%) | -0.017 | 728 (33.6%) | 754 (34.8%) | -0.025 |
| Other rheumatic disorders (including gout); n (%)* | 550 (73.6%) | 548 (73.4%) | 0.005 | 997 (70.2%) | 1,005 (70.8%) | -0.017 | 1,547 (71.4%) | 1,553 (71.7%) | -0.023 |
| | | | 0.003 | | | 0.000 | | | 0.022 |
| Gout and other crystal arthropathies; n (%) | 21 (2.8%) | 15 (2.0%) | | 25 (1.8%) | 25 (1.8%) | | 046 (2.1%) | 040 (1.8%) | |
| Other rheumatic disorders; n (%)* | 547 (73.2%) | 546 (73.1%) | 0.002 | 991 (69.8%) | 1,000 (70.4%) | -0.013 | 1,538 (71.0%) | 1,546 (71.3%) | -0.007 |
| Neuro Conditions | | | | | | | | | |
| Parkinson's disease; n (%) | 1 (0.1%) | 0 (0.0%) | 0.045 | 3 (0.2%) | 1 (0.1%) | 0.026 | 004 (0.2%) | 001 (0.0%) | 0.063 |
| Alzheimer and other Dementia Disease ; n (%)* | 49 (6.6%) | 56 (7.5%) | -0.035 | 71 (5.0%) | 86 (6.1%) | -0.048 | 120 (5.5%) | 142 (6.6%) | -0.046 |
| Seizure disorders (epilepsy); n (%) | 17 (2.3%) | 13 (1.7%) | 0.043 | 26 (1.8%) | 27 (1.9%) | -0.007 | 043 (2.0%) | 040 (1.8%) | 0.015 |
| Delirium/Psychosis; n (%) | 30 (4.0%) | 31 (4.1%) | -0.005 | 35 (2.5%) | 57 (4.0%) | -0.085 | 065 (3.0%) | 088 (4.1%) | -0.059 |
| Other Conditions | | | | | | | | | |
| Vitamin D deficiency; n (%)* | 212 (28.4%) | 206 (27.6%) | 0.018 | 218 (15.4%) | 217 (15.3%) | 0.003 | 430 (19.8%) | 423 (19.5%) | 0.008 |
| Liver disease; n (%)* | 26 (3.5%) | 33 (4.4%) | -0.046 | 49 (3.5%) | 47 (3.3%) | 0.011 | 075 (3.5%) | 080 (3.7%) | -0.011 |
| Chronic kidney disease stages I-III; n (%)* | 70 (9.4%) | 74 (9.9%) | -0.017 | 65 (4.6%) | 59 (4.2%) | 0.020 | 135 (6.2%) | 133 (6.1%) | 0.004 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 21 (2.8%) | 17 (2.3%) | 0.032 | 18 (1.3%) | 21 (1.5%) | -0.017 | 039 (1.8%) | 038 (1.8%) | 0.000 |
| Premature menopause; n (%) | 1 (0.1%) | 3 (0.4%) | -0.060 | 1 (0.1%) | 1 (0.1%) | 0.000 | 002 (0.1%) | 004 (0.2%) | -0.026 |
| Oophorectomy; n (%) | 1 (0.1%) | 0 (0.0%) | 0.045 | 0 (0.0%) | 1 (0.1%) | -0.045 | 001 (0.0%) | 001 (0.0%) | 0.000 |
| COPD; n (%)* | 123 (16.5%) | 130 (17.4%) | -0.024 | 214 (15.1%) | 207 (14.6%) | 0.014 | 337 (15.6%) | 337 (15.6%) | 0.000 |
| Asthma; n (%)* | 80 (10.7%) | 88 (11.8%) | -0.035 | 132 (9.3%) | 135 (9.5%) | -0.007 | 212 (9.8%) | 223 (10.3%) | -0.017 |
| Obstructive sleep apnea; n (%)* | 49 (6.6%) | 48 (6.4%) | 0.008 | 56 (3.9%) | 50 (3.5%) | 0.021 | 105 (4.8%) | 098 (4.5%) | 0.017 |
| Syncope; n (%)* | 39 (5.2%) | 45 (6.0%) | -0.035 | 77 (5.4%) | 85 (6.0%) | -0.026 | 116 (5.4%) | 130 (6.0%) | -0.026 |
| Falls; n (%)* | 134 (17.9%) | 142 (19.0%) | -0.028 | 79 (5.6%) | 81 (5.7%) | -0.004 | 213 (9.8%) | 223 (10.3%) | -0.017 |
| VTE; n (%) | 33 (4.4%) | 32 (4.3%) | 0.005 | 49 (3.5%) | 47 (3.3%) | 0.011 | 082 (3.8%) | 079 (3.6%) | 0.011 |
| Gait abnormality; n (%)* | 141 (18.9%) | 140 (18.7%) | 0.005 | 167 (11.8%) | 166 (11.7%) | 0.003 | 308 (14.2%) | 306 (14.1%) | 0.003 |
| Osteopenia; n (%)* | 256 (34.3%) | 247 (33.1%) | 0.025 | 316 (22.3%) | 315 (22.2%) | 0.002 | 572 (26.4%) | 562 (25.9%) | 0.011 |
| History of hip and femur fractures; n (%)* | 41 (5.5%) | 45 (6.0%) | -0.021 | 105 (7.4%) | 102 (7.2%) | 0.008 | 146 (6.7%) | 147 (6.8%) | -0.004 |
| Other Fractures ; n (%)* | 90 (12.0%) | 95 (12.7%) | -0.021 | 170 (12.0%) | 160 (11.3%) | 0.022 | 260 (12.0%) | 255 (11.8%) | 0.006 |
| Glucocorticoid-Induced Osteoporosis; n (%)* | 2 (0.3%) | 2 (0.3%) | 0.000 | 1 (0.1%) | 2 (0.1%) | 0.000 | 003 (0.1%) | 004 (0.2%) | -0.026 |
| Combined comorbidity score | | | | | | | | | |
| mean (sd) | 1.20 (2.17) | 1.25 (2.25) | -0.023 | 0.90 (1.71) | 0.86 (1.72) | 0.023 | 1.00 (1.88) | 0.99 (1.92) | 0.005 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.000 | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.000 | 0.34 (1.88) | 0.34 (1.92) | 0.000 |
| Frailty Score: Empirical Version 365 days as Categories | | | | | | | | | |
| <0.12908; n (%) | 317 (42.4%) | 318 (42.6%) | -0.004 | 476 (33.5%) | 472 (33.2%) | 0.006 | 793 (36.6%) | 790 (36.5%) | 0.002 |
| 0.12908 - 0.1631167; n (%) | 158 (21.2%) | 155 (20.7%) | 0.012 | 309 (21.8%) | 318 (22.4%) | -0.014 | 467 (21.6%) | 473 (21.8%) | -0.005 |
| >= 0.1631167; n (%) | 272 (36.4%) | 274 (36.7%) | -0.006 | 635 (44.7%) | 630 (44.4%) | 0.006 | 907 (41.9%) | 904 (41.7%) | 0.004 |
| Medication Use | , , | , , | | , , | , , | | , , | , , | |
| Use of oral corticosteroids; n (%)* | 268 (35.9%) | 266 (35.6%) | 0.006 | 498 (35.1%) | 506 (35.6%) | -0.010 | 766 (35.3%) | 772 (35.6%) | -0.006 |
| Use of antidepressants; n (%)* | 256 (34.3%) | 275 (36.8%) | -0.052 | 606 (42.7%) | 576 (40.6%) | 0.043 | 862 (39.8%) | 851 (39.3%) | 0.010 |
| Use of anticonvulsants; n (%)* | 159 (21.3%) | 149 (19.9%) | 0.035 | 323 (22.7%) | 311 (21.9%) | 0.019 | 482 (22.2%) | 460 (21.2%) | 0.024 |
| Use of beta blocker OR calcium channel blocker; n (%)* | 250 (33.5%) | 235 (31.5%) | 0.033 | 471 (33.2%) | 478 (33.7%) | -0.011 | 721 (33.3%) | 713 (32.9%) | 0.009 |
| Use of PPIs; n (%)* | 222 (29.7%) | 219 (29.3%) | 0.009 | 488 (34.4%) | 501 (35.3%) | -0.019 | 710 (32.8%) | 720 (33.2%) | -0.009 |
| Use of opioids; n (%)* | 419 (56.1%) | 420 (56.2%) | -0.002 | 848 (59.7%) | 853 (60.1%) | -0.008 | 1,267 (58.5%) | 1,273 (58.7%) | -0.004 |
| Use of antipsychotics; n (%)* | 21 (2.8%) | 24 (3.2%) | -0.023 | 53 (3.7%) | 54 (3.8%) | -0.005 | 074 (3.4%) | 078 (3.6%) | -0.011 |
| Use of anxiolytics/hypnotics; n (%)* | 74 (9.9%) | 88 (11.8%) | -0.061 | 249 (17.5%) | 228 (16.1%) | 0.037 | 323 (14.9%) | 316 (14.6%) | 0.008 |
| Use of dementia meds; n (%)* | 34 (4.6%) | 32 (4.3%) | 0.015 | 73 (5.1%) | 69 (4.9%) | 0.009 | 107 (4.9%) | 101 (4.7%) | 0.009 |
| Use of antiparkinsonian meds; n (%)* | 21 (2.8%) | 26 (3.5%) | -0.040 | 58 (4.1%) | 64 (4.5%) | -0.020 | 079 (3.6%) | 090 (4.2%) | -0.031 |
| Use of Benzodiazepine; n (%)* | 146 (19.5%) | 162 (21.7%) | -0.054 | 404 (28.5%) | 382 (26.9%) | 0.036 | 550 (25.4%) | 544 (25.1%) | 0.007 |
| All antidiabetic medications; n (%)* | 78 (10.4%) | 73 (9.8%) | 0.020 | 162 (11.4%) | 166 (11.7%) | -0.009 | 240 (11.1%) | 239 (11.0%) | 0.003 |
| ACEI/ARB; n (%)* | 261 (34.9%) | 256 (34.3%) | 0.013 | 470 (33.1%) | 475 (33.5%) | -0.008 | 731 (33.7%) | 731 (33.7%) | 0.000 |
| Use of Anticoagulants; n (%)* | 71 (9.5%) | 72 (9.6%) | -0.003 | 158 (11.1%) | 148 (10.4%) | 0.023 | 229 (10.6%) | 220 (10.2%) | 0.013 |
| Use of Amiodarone; n (%) | 9 (1.2%) | 8 (1.1%) | 0.009 | 19 (1.3%) | 23 (1.6%) | -0.025 | 028 (1.3%) | 031 (1.4%) | -0.009 |
| 1 | | - 11 | | - / | - (=/ | | (/ | , , | |

| | 1 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Digoxin; n (%) | 18 (2.4%) | 14 (1.9%) | 0.034 | 45 (3.2%) | 38 (2.7%) | 0.030 | 063 (2.9%) | 052 (2.4%) | 0.031 |
| Use of Diuretics; n (%)* | 205 (27.4%) | 220 (29.5%) | -0.047 | 466 (32.8%) | 466 (32.8%) | 0.000 | 671 (31.0%) | 686 (31.7%) | -0.015 |
| Use of Aspirin; n (%) | 5 (0.7%) | 5 (0.7%) | 0.000 | 25 (1.8%) | 24 (1.7%) | 0.008 | 030 (1.4%) | 029 (1.3%) | 0.009 |
| NSAIDs (NOT including aspirin); n (%) | 203 (27.2%) | 188 (25.2%) | 0.045 | 377 (26.5%) | 318 (22.4%) | 0.096 | 580 (26.8%) | 506 (23.4%) | 0.078 |
| HRT (Use of estrogens, progestins, androgens); n (%)* | 47 (6.3%) | 44 (5.9%) | 0.017 | 84 (5.9%) | 93 (6.5%) | -0.025 | 131 (6.0%) | 137 (6.3%) | -0.012 |
| Other Pressors; n (%) | 5 (0.7%) | 5 (0.7%) | 0.000 | 8 (0.6%) | 20 (1.4%) | -0.080 | 013 (0.6%) | 025 (1.2%) | -0.064 |
| Use of Statins ; n (%)* | 258 (34.5%) | 252 (33.7%) | 0.017 | 521 (36.7%) | 523 (36.8%) | -0.002 | 779 (35.9%) | 775 (35.8%) | 0.002 |
| Selective Estrogen Receptor Modulators (SERMs); n (%)* | 7 (0.9%) | 19 (2.5%) | -0.124 | 31 (2.2%) | 38 (2.7%) | -0.032 | 038 (1.8%) | 057 (2.6%) | -0.055 |
| Healthcare Utilization Measures | | | | | | | | | |
| Use of any drugs claims* | | | | | | | | | |
| mean (sd) | 24.76 (18.01) | 24.95 (18.56) | -0.010 | 25.89 (19.03) | 25.43 (18.22) | 0.025 | 25.50 (18.68) | 25.26 (18.34) | 0.013 |
| Number of office visits* | | | | | | | | | |
| mean (sd) | 11.57 (7.84) | 11.48 (7.34) | 0.012 | 11.99 (8.51) | 11.90 (7.78) | 0.011 | 11.85 (8.29) | 11.76 (7.63) | 0.011 |
| Number of ED visits* | | | | | | | | | |
| mean (sd) | 0.69 (1.22) | 0.76 (1.17) | -0.059 | 0.59 (1.19) | 0.60 (1.22) | -0.008 | 0.62 (1.20) | 0.66 (1.20) | -0.033 |
| Number of Hospitalizations* | | | | | | | | | |
| mean (sd) | 0.46 (1.02) | 0.46 (1.02) | 0.000 | 2.09 (5.83) | 2.09 (5.52) | 0.000 | 1.53 (4.76) | 1.53 (4.51) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 14 (1.9%) | 19 (2.5%) | -0.041 | 28 (2.0%) | 29 (2.0%) | 0.000 | 042 (1.9%) | 048 (2.2%) | -0.021 |
| Old hospitalizations (-450 to -31 days); n (%) | 163 (21.8%) | 167 (22.4%) | -0.014 | 356 (25.1%) | 360 (25.4%) | -0.007 | 519 (24.0%) | 527 (24.3%) | -0.007 |
| Number of Endocrinologist visits* | , | . , | | , | , , | | , | , | |
| mean (sd) | 0.41 (1.19) | 0.43 (1.11) | -0.017 | 1.75 (2.89) | 1.73 (2.94) | 0.007 | 1.29 (2.44) | 1.28 (2.47) | 0.004 |
| Number of DXA test performed* | , , , | , | | . , , | - ( - / | | , | - ( , | |
| mean (sd) | 0.73 (0.63) | 0.73 (0.54) | 0.000 | 0.49 (0.52) | 0.49 (0.52) | 0.000 | 0.57 (0.56) | 0.57 (0.53) | 0.000 |
| Number of hospital days* | J | (0.0) | | (0.02) | ( ) | | () | | |
| mean (sd) | 5.18 (17.50) | 4.98 (17.59) | 0.011 | 2.09 (5.83) | 2.09 (5.52) | 0.000 | 3.16 (11.30) | 3.09 (11.25) | 0.006 |
| Occurrence of basic or comprehensive blood chemistry test; n (%)* | 577 (77.2%) | 573 (76.7%) | 0.012 | 626 (44.1%) | 615 (43.3%) | 0.016 | 1,203 (55.5%) | 1,188 (54.8%) | 0.014 |
| Number of HbA1C test ordered* | 377 (77.1270) | 373 (70.770) | 0.012 | 020 (11.270) | 015 (15.570) | 0.010 | 1,200 (00.070) | 1,100 (5 1.070) | 0.01 |
| mean (sd) | 0.55 (1.09) | 0.54 (1.15) | 0.009 | 0.27 (0.78) | 0.26 (0.79) | 0.013 | 0.37 (0.90) | 0.36 (0.93) | 0.011 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%)* | 64 (8.6%) | 68 (9.1%) | -0.018 | 142 (10.0%) | 138 (9.7%) | 0.010 | 206 (9.5%) | 206 (9.5%) | 0.000 |
| Number of Mammograms (Breast cancer screening); n (%)* | 352 (47.1%) | 359 (48.1%) | -0.020 | 547 (38.5%) | 545 (38.4%) | 0.002 | 899 (41.5%) | 904 (41.7%) | -0.004 |
| Number of Pap smear (Cervical cancer screening); n (%)* | 144 (19.3%) | 138 (18.5%) | 0.020 | 264 (18.6%) | 265 (18.7%) | -0.003 | 408 (18.8%) | 403 (18.6%) | 0.005 |
| Flu vaccine; n (%)* | 278 (37.2%) | 273 (36.5%) | 0.020 | 312 (22.0%) | 314 (22.1%) | -0.003 | 590 (27.2%) | 587 (27.1%) | 0.003 |
| Pneumococcal vaccine; n (%)* | 132 (17.7%) | 135 (18.1%) | -0.010 | 125 (8.8%) | 134 (9.4%) | -0.002 | 257 (11.9%) | 269 (12.4%) | -0.015 |
| Copay for pharmacy cost (charges in U.S. \$)* | 132 (17.7%) | 133 (10.1%) | -0.010 | 123 (8.8%) | 134 (9.4%) | -0.021 | 237 (11.3%) | 209 (12.4%) | -0.015 |
| mean (sd) | 36.14 (46.87) | 34.80 (42.78) | 0.030 | 21.56 (22.23) | 21.55 (23.62) | 0.000 | 26.59 (32.88) | 26.12 (31.56) | 0.015 |
| * * | , , | , , | | , , | , , | -0.005 | , , | . , | |
| median [IQR] | 23.44 [13.37, 42.35]<br>NA | 25.00 [11.82, 41.43] | -0.035 | 17.18 [7.87, 29.33]<br>NA | 17.29 [8.09, 28.68]<br>NA | | 19.34 (32.88) | 19.95 (31.56) | -0.019<br>NA |
| Missing; n (%) | NA NA | NA | NA | NA | NA NA | NA | NA | NA | NA |
| Business Type* | 224 (22 224) | 204 (20 204) | | | | | 204 (20 204) | 204 (20 004) | |
| Commercial; n (%) | 291 (39.0%) | 291 (39.0%) | 0.000 | NA<br> | NA | NA | 291 (39.0%) | 291 (39.0%) | 0.000 |
| Medicare; n (%) | 456 (61.0%) | 456 (61.0%) | 0.000 | NA | NA | NA | 456 (61.0%) | 456 (61.0%) | 0.000 |
| Insurance Plan Type* | | | | | | | | | |
| Comprehensive; n (%) | NA | NA | NA | 413 (29.1%) | 431 (30.4%) | -0.028 | 413 (29.1%) | 431 (30.4%) | -0.028 |
| HMO; n (%) | NA | NA | NA | 97 (6.8%) | 104 (7.3%) | -0.020 | 97 (6.8%) | 104 (7.3%) | -0.020 |
| PPO; n (%) | NA | NA | NA | 731 (51.5%) | 705 (49.6%) | 0.038 | 731 (51.5%) | 705 (49.6%) | 0.038 |
| Others; n (%) | NA | NA | NA | 179 (12.6%) | 180 (12.7%) | -0.003 | 179 (12.6%) | 180 (12.7%) | -0.003 |

<sup>\*</sup>Included in the 1:1 PS matching model